### Intranasal dexmedetomidine for laceration repair in children: a dose finding study

### **Trial registration:**

Clinicaltrials.gov Identified Number: NCT03957304

Protocol number: DFS05081977

Protocol Version Number: V 3.5, 2019-11-01

### **Funding:**

Children's Health Research Institute and Lawson Internal Research Fund. The funders have no role or authority in study design, collection, management, analysis, and interpretation of data, writing of the report, or the decision to submit the report for publication.

### **Study Sponsor:**

Dr. Naveen Poonai, MSc MD FRCPC

Associate Professor of Pediatrics & Internal Medicine

Schulich School of Medicine & Dentistry

Associate Scientist, Child Health Research Institute Research Director

Division of Paediatric Emergency Medicine

800 Commissioners Road East, Room E1-106, London, Ontario, N6A 5W9

Phone: 519 694 5309/ Fax: 519 667 6769 Alternate email: naveen.poonai@lhsc.on.ca

### **Qualified Principal Investigator:**

Dr. Naveen Poonai

#### **Co-Investigators (Name and Department):**

- Dr. Vikram Sabhaney, MD, Assistant Professor, Paediatrics, University of British Columbia
- Dr. Samina Ali, MDCM, Professor, Paediatrics, University of Alberta
- Dr. Kamary Coriolano, PhD, Clinical Research Coordinator, London Health Sciences Centre
- Dr. Maala Bhatt, MD, Associate Professor, Paediatrics, University of Ottawa
- Dr. Evelyne Doyon-Trottier, MD, Associate Professor, Paediatrics, Universite de Montreal
- Dr. Amit Shah, MD, Associate Professor, Internal Medicine, Western University
- Dr. Anna Heath, PhD, The Hospital for Sick Children, Assistant Professor

### **Collaborators:**

Ms. Kyna Patterson, Child Life Specialist, London Health Sciences Centre

### **Roles and Responsibilities:**

Dr. Poonai is the lead investigator responsible for trial oversight. Dr. Coriolano is the project coordinator. Dr. Heath is the biostatistician responsible for data analysis. All other investigators

are knowledge experts that will contribute to the design, protocol, results interpretation, and manuscript preparation.

### **INTRODUCTION**

### Lay Summary

The most common injury prompting an emergency department (ED) visit in children is a cut (laceration) that requires repair using stitches or skin glue. Despite anesthetic (freezing), laceration repair is often very distressful because in young children, most occur on the face. Distraction techniques are difficult and restraint is often necessary to achieve a cosmetically appealing repair. Although pain can usually be minimized, distress is very difficult to manage in children. Drugs to reduce anxiety in adults such as lorazepam (Ativan<sup>TM</sup>) often produce greater anxiety in children. There is currently no effective drug to relieve the distress of laceration repair in children. Untreated pain and distress in children results in slower healing, poor appetite and sleep, fear of medical care, and chronic pain. Parents are significantly affected by witnessing their child's discomfort and look to health providers to relieve pain and distress. Our goal is to find a safe and effective drug to reduce distress in children undergoing laceration repair. Dexmedetomidine is a new drug that safely provides mild sedation and can be given as a painless nasal spray. Intranasal dexmedetomidine (IND) has been shown to reduce distress in children undergoing painful procedures such as dental work and intravenous insertion. However, no large study has explored IND for laceration repair. In order for research to change the way we care for children, a large study that enrolls children across many paediatric EDs needs to be performed. The first step is to conduct a smaller study to identify the safest and most effective dose. Our proposed study plans to enroll 55 children age 1-10 years who require laceration repair. Each participant will receive a weight-based dose of IND with 1-2 pairs of nasal sprays. Different doses will be used until the most effective and safe dose is found. All children will receive local anesthetic (freezing) and undergo laceration repair according to standard practice. The two most important outcomes during the procedure are sedation and anxiety. We will record a video of the child during laceration repair and to reduce bias, videos will be scored by research assistants who are not in the ED. The parent, child, nurse, and doctor will rate their satisfaction with the procedure using a 5-point scale. Following discharge, at 24-48 hours, the family will receive a 10-minute Internet-based survey to identify delayed adverse behaviors and at 14 days, a 3-minute survey to record complications related to laceration repair. Our results will be used to design a larger study which may potentially lead to a much less distressing experience for children that require laceration repair. Perceived distress in children is closely tied to caregiver satisfaction and an improved ED experience will lead to a more positive view of the health care team. A more relaxed child will enhance the ability of doctors and trainees to achieve a good cosmetic repair. Given our links with surrounding hospitals where most children with lacerations attend, our results can easily be shared to improve the care of children across Southwestern Ontario and eventually Canada-wide.

### **Background and Rationale**

Lacerations are the most common injury for which children seek care in the emergency department (ED) (1). In Canada, lacerations are one of the top ten presenting complaints in

children under 10 years, comprising nearly 8% of paediatric ED visits (2). Despite the routine application of topical lidocaine-epinephrine-tetracaine (LET) for analgesia, young children routinely resist laceration repair. While distraction may help in older children, in younger children, most lacerations occur on the face (3), making distraction difficult. Untreated pain in childhood can lead to short-term problems such as slower healing and long-term issues such as anxiety, needle phobia, and fear of medical care as adults (4). In 2016, the American Academy of Pediatrics and American Academy of Pediatric Dentistry recommended a goal of minimizing discomfort and pain and controlling behavior and movement during procedures (5). Local or topical anesthetics may reduce pain but do nothing to alleviate procedural distress (6). Many children require light sedation to provide comfort, promote compliance with positioning requirements, and facilitate a timely and cosmetically appealing repair (6). Intranasal midazolam is the most commonly used anxiolytic in children, however, a systematic review found little evidence of benefit (7). Moreover, midazolam has unpredictable efficacy and discomfort with nasal administration is a common complaint (8, 9). Dexmedetomidine is a relatively new alpha-2adrenergic receptor agonist with anxiolytic, sedative, and analgesic properties (10). Three systematic reviews have suggested intravenous dexmedetomidine is effective for procedural distress in children (10-12). However, intranasal therapies are gaining popularity among health care providers due to ease of administration and less distress. Consequently, our team performed a systematic review of intranasal dexmedetomidine (IND). The review included 18 trials of 2037 children undergoing distressing procedures including intravenous insertion, dental extraction, ophthalmologic examination, and diagnostic imaging (Appendix A). Across trials, IND had an onset and duration of sedation of 7-31 and 41-92 minutes, respectively. IND 1-4 mcg/kg provided adequate sedation in a significantly greater proportion of children (79%, range 55-98%) versus other anxiolytics (midazolam, chloral hydrate) (60%, range 0-96%). There were no serious adverse events and IND was well tolerated in 88% of participants (13). However, heterogeneity in dose and vehicle (mucosal atomizer versus nasal drops) underscored the wide range in effectiveness we observed. Optimizing these factors may produce more consistent and effective sedation. Due to heterogeneity, we were unable to characterize a dose-response relationship and an area of uncertainty is the optimal dose of IND. Only one trial has investigated IND in children for positioning prior to laceration repair. 70% (n=20) of participants were deemed "not anxious" compared to intranasal midazolam (11%, n=18) (3). However, the small sample size and focus on pre-procedural anxiety have limited clinical uptake. A large multicentre trial with an optimized dosing protocol will yield the best estimate of IND's effectiveness. The results will be more likely to improve how the distress of laceration repair is managed. However, this is predicated upon determining recruitment feasibility, protocol compliance, and the most effective dose of IND.

### Purpose of the study

Currently, an effective drug to relieve the distress of laceration repair in children is not known. Therefore, purpose of this study is to find a safe and effective drug to reduce distress in children undergoing laceration repair.

### **Expected Results and Significance**

We believe that our study will identify the most efficacious and safe dose of IND, logistic obstacles to recruitment, and a realistic expectation of maximal sedation efficacy. The results will

inform the design of a much larger multicentre randomized trial that will hopefully change practice and improve care.

### **Objectives**

### **Primary Objective:**

In children aged 1 to 10 years who requires a laceration repair using stitches or skin glue, our objective is to determine the most efficacious dose of intranasal dexmedetomidine (IND) in terms of adequate sedation for laceration repair. Adequate sedation for the duration of the laceration repair is measured using the Pediatric Sedation State Scale (PSSS) (14).

### Secondary Objectives:

- 1. To determine how well participants were able to tolerate the IND sprays.
- 2. To determine the degree of satisfaction with laceration repair on the part of participants and health care providers
- 3. To determine the feasibility of recruitment
- 4. To determine the logistic obstacles to implementation

We hypothesize that adequate sedation will be seen at higher doses of IND (3-4 mcg/kg) compared to lower doses (1-2 mcg/kg). Our objectives are to determine: (i) the most efficacious dose of IND in terms of adequate sedation for laceration repair, (ii) tolerability of IND sprays, (iii) patient and provider satisfaction with laceration repair, (iv) feasibility of recruitment, (v) logistic obstacles to implementation

### Limitations

Scoring of sedation and anxiolysis are subjective which may lead to an inaccurate determination of the optimal dose. To minimize this risk, the training protocol used in prior studies employing the PSSS will be followed. In addition, a kappa statistic < 0.7 will prompt a re-review of the videos by the PI. Blinding of the different doses will be difficult to accomplish and may be a source of bias. To overcome this, the outcome assessors scoring the videos for sedation (PSSS) and anxiety (YPAS) will be remote from the clinical encounter and the video segment will commence following intranasal drug administration.

### **Trial Design**

This study will be designed as a phase II single-arm dose ranging pilot study using an adapted version of the Continual Reassessment Method (15). CRM is a model-based design that is more likely to determine the correct dose compared to standard 3+3 designs (16). The adapted method adjusts for potential over-sedation (as measured by the PSSS) for higher doses of IND.

### METHODS: PARTICIPANTS, INTERVENTIONS, AND OUTCOMES

### **Study Setting**

This study will be carried out in the paediatric emergency department (ED) of the Children's Hospital in London, Ontario, Canada.

### Eligibility criteria

### Inclusion Criteria

We will **include** (i) children age 1-10 years who present to the ED with a single isolated laceration ≤ 5 cm deemed to require single-layer closure using sutures based on the opinion of the treating physician, (ii) predicted to resist positioning for laceration repair based on the opinion of the caregiver, treating physician, child life specialist, or bedside nurse, (iii) lidocaine/epinephrine/tetracaine (LET) used as sole initial topical anesthetic agent

### **Exclusion Criteria**

We will exclude children with (i) laceration repair requiring procedural sedation (without IND) or local nerve block, (ii) other injuries requiring reduction (fracture or dislocation) or repair (nailbed injury or laceration), (iii) lacerations containing foreign body material (including dirt and debris), (iv) history of hypersensitivity to dexmedetomidine, (v) occlusion of at least one nare due to mucus, polyps, septal deviation, etc., (vi) concomitant use of an a2-adrenergic receptor agonist, (vii) bradycardia or hypotension for age (possible transient but clinically insignificant adverse effects of dexmedetomidine), (viii) we will exclude caregivers if they are not the primary care provider, (ix) are unable to read or understand English above at least a grade 8 literacy level, (x) concomitant upper respiratory tract infection or allergic rhinitis with at least one non-patent nare, (xi) known renal insufficiency, (xii) uncorrected mineralocorticoid deficiency, (xiii) congenital heart disease or cardiac conduction disorder

### Intervention

### **Description of intervention**

Participants will be consecutively screened for eligibility during the hours of study recruitment (1700 to 2300 hours, 7 days per week) by trained research assistants (RA) prior to being seen by a physician but after nursing assessment. If eligible, the RA will obtain informed consent and assent (when applicable) and the physician will confirm eligibility and order the study intervention on Cerner. Participants will be administered IND 100 mcg/mL [Precedex®, Pfizer Canada Inc, Kirkland, Québec 1-4 mcg/kg (max 200 mcg or 2 mL)]. The weight-based dose will be calculated by REDCap and confirmed by the nurse and physician. The intervention will be drawn into a mucosal atomizer device (MAD) by the bedside nurse using a 1 mL syringe. An extra 0.15 mL will be drawn into the atomizer upon first use to account for dead space. No more than 0.5 mL per nare will be administered at once because volumes exceeding 0.5 mL result in oropharyngeal deposition (17). If two sprays are required (one per nare), they will be administered either simultaneously or in rapid succession. IND will be administered by the bedside nurse with the participant positioned supine with the head at 45°. In our ED, topical anesthetic (LET) is placed on the wound 30 minutes prior to laceration repair once the nurse has obtained a physician's order. IND has a time to peak plasma concentration of 38 minutes (17) and an onset of sedation in children of 25 minutes (18). IND will be given at the same time as LET placement so that the onset of sedation is coincident with positioning for laceration repair. The physician or their designate will be asked to perform suture repair after at least 30 minutes has elapsed following IND administration.

The RA will conduct two follow-ups with participants by email or telephone, depending on the preference of the participant. The RA will contact the participant 24-48 hours post-discharge to identify the presence of delayed maladaptive behaviors using the Post-Hospital Behavior Questionnaire (PHBQ); The PHBQ will take approximately 10 minutes to complete. At 14 days post-laceration repair, participants will be contacted to determine the presence or absence of complications (infection; dehiscence; contracture; retained suture material). This survey will take approximately 3 minutes to complete. If the latter survey cannot be obtained, the medical record of the participant will be examined for the presence of an emergency department visit for wound-related complications.

### Criteria for discounting or modifying allocated interventions

An investigator may discontinue or withdraw a participant from the study for the following reasons:

- 1. If any clinical adverse event (AE), laboratory abnormality, or other medical condition or situation occurs such that continued participation in the study would be detrimental to the health of the participant.
- 2. If the participant is found to meet exclusion criteria (either newly developed or not previously recognized) that precludes further study participation.

### Concomitant care and interventions that are permitted or prohibited during the trial

Permissible co-interventions include topical and subcutaneous anesthetic, oral or IV analgesics, and non-pharmacologic strategies for pain and distress.

### **Outcomes**

All data will be recorded using Research Electronic Data Capture (REDCap) by RAs. We will collect demographic data: age; sex; size and location of laceration; number of sutures; trainee level (if repair is not performed by attending physician); type of local anesthetic; presence or absence of a child life specialist; distraction techniques; data pertaining to primary and secondary outcomes. The **primary outcome** is adequate sedation (PSSS 2 or 3) for the duration of the measurement period (initial positioning to tying of the last suture). **Secondary outcomes** include: onset and duration of sedation; adverse effects as defined by the Quebec Guidelines (16); anxiolysis during the study period measured using the *Yale Preoperative Anxiety Scale*; compliance (yes/no) with IND administration; satisfaction with laceration repair using a 5-item Likert scale obtained from the caregiver, child (if > 7 years), individual performing the repair, and bedside nurse; nasal irritation from children age > 4 years using the *Faces Pain Scale – Revised* (FPS-R); length of stay; consent rate; heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP) and oxygen saturation (SpaO2), respiratory rate (RR) recorded at baseline and every 5 minutes until 60 minutes after last pair of sprays is administered, delayed maladaptive behaviors using the *Post-Hospital Behavior Questionnaire* (PHBQ) assessed 24-48 hours post

discharge; complications within 14 days of discharge (infection; dehiscence; contracture; retained suture material).

### **Patient Engagement**

Study outcomes were identified and agreed upon by a five-member focus group involving the PI, a child life specialist, and three parents of children who have undergone laceration repair. The study design therefore reflects their concerns about length of stay and topical analgesia.

### **Participant timeline**



Study: Intranasal dexmedetomidine for laceration repair in children: a dose finding study

Protocol: Dose Finding Study Version 3.5 – November 1, 2019

### Sample Size

This was calculated using the *Bayesian Continual Reassessment Method* (18). Based on an adverse event rate of 20%, an "effect size" of 1.6 (i.e. the odds ratio between consecutive increasing doses), and a phase II trial accuracy level of 60%, we estimated a sample size of 50 participants. With increasing the sample size by 10% to account for dropouts, the final sample size is 55 participants.

### **Feasibility**

An existing team of 12 research assistants (RAs) with REDCap and clinical trial recruitment experience are available to recruit during the peak visit period of 1700-2300 hours, 7 days a week, 50 weeks a year. A 2018 clinical informatics search revealed that 1332 laceration repairs were performed, of which 472 met our inclusion criteria and presented between 1700-2300 hours. With an expected 50% consent rate, recruitment of 50 participants is feasible in 12 months.

#### Recruitment

**METHODS: ASSIGNMENT OF INTERVENTIONS** 

### **Allocation**

Not applicable

### **Sequence generation**

A list will be provided to

### Allocation concealment mechanism

Not applicable

### **Implementation**

Participants will be assigned to each dosing level by pharmacy based on the continual reassessment method's study design. Research assistants will enroll participants.

### **Blinding**

Blinding of dose levels will not be possible for clinical and research personnel in the ED. However, outcome assessors will be blinded by virtue of being remote from the clinical encounter. Furthermore, video segments will commence immediately after intranasal sprays are given so outcome assessors will not see what volume is administered. Two independent assessors will score each video and an inter-rater agreement (kappa) will be calculated. Disagreements on

scoring for the purposes of estimating the Bayesian dose response model will be resolved by discussion.

### METHODS: DATA COLLECTION, MANAGEMENT, AND ANALYSIS

#### **Data collection methods**

Sedation will be measured using the Pediatric Sedation State Scale (PSSS) (Appendix B), an instrument validated for video scoring of children undergoing painful procedures. The PSSS is scored from 0 to 5 easily by non-medical personnel. The PSSS assesses pain as well as over sedation and under sedation. Adequate sedation is a score of 2 or 3, over sedation is a score of 0 or 1 and under sedation is a score of 4 or 5 (14). Participants will be assigned to doses of IND from 1-4 mcg/kg, increasing in whole number increments. Initially three participants will receive 1mcg/kg and the number of participants at each dose of IND will be recorded. Data from these participants will be used to update a Bayesian model for the dose-response curve for all three categories of sedation. The following three participants will be assigned the dose with the highest posterior probability of an efficacy close to 0.8. This balances the need to determine the most efficacious dose but prevents an excessive number of over-sedations. For the Bayesian dose response model, a determination will be made as to the overall score category for each participant ("adequate", "over", or "under sedated" based on the PSSS). To be scored as "adequate", a participant must have a PSSS score of 2 or 3 for at least 90% of observations from initial positioning to tying of the last suture. If a participant does not retain a PSSS score of 2 or 3 for at least 90% of the observations, they will be categorized as either over or under-sedated, if the majority of the remaining PSSS scores are 0 or 1 or 4 or 5, respectively. Furthermore, if the participant remains awake, but not distressed during the procedure, they will be scored as a 2 based on the PSSS. However, for the purposes of the Bayesian dose response model, they will be scored as "under sedated" to avoid concluding that a lower dose of IND is effective based on the outcomes for participants that did not require sedation. Finally, participants who are noncompliant with IND will be categorized as an over-sedation as it is assumed that this dose was not well tolerated by the participant and dose escalation should be avoided.

Preliminary results indicate that, conditional on suitable priors, this method has an approximately 83% chance of selecting the most effective dose. Serious adverse events as defined by the Quebec Guidelines on paediatric procedural sedation (19) will be reported as per Good Clinical Practices. Data will be reviewed after each dose by a data safety monitoring board (DSMB), who will confirm it is safe to escalate to the dose proposed using the Bayesian dose response model. The DSMB will be comprised of two emergency physicians and will be independent from the sponsor and reporting structure. Permissible co-interventions include topical and subcutaneous anesthetic, oral or IV analgesics, and non-pharmacologic strategies for pain and distress.

### **Data management**

The site investigator will be responsible for retaining (archiving) their own essential study documents that individually or collectively permit the evaluation and conduct of the study and the

quality of data, in accordance with ICH-GCP and applicable regulatory requirements. All study documents, including source, are to be stored in a confidential location with secured and limited access. All electronic records and data sets will be encrypted and password protected with access only permitted by the PI, site coordinator(s), and research team members. Paper data (e.g. copies of consent and assent forms) will be stored exclusively in the Participating Site Investigator's research office in a locked cabinet. Results will not be reported in a way that identifies any individuals.

All study related documentation will be retained in accordance with Health Canada's Food and Drug Regulations for 25 years and per the investigational site's institutional record management and retention policies. No records will be destroyed without the written consent of the Qualified Investigator and/or Sponsor.

### **Statistical methods**

For demographic data and all secondary outcomes, we will summarize the data using

- i) proportions for discrete variables
- ii) means, medians, standard deviation, interquartile range and range for continuous variables For the primary outcome, we will also provide the Bayesian credible interval for the probability of a successful sedation, estimated from the Bayesian dose response curve. We will provide a graphical summary of patient flow and the dose escalation process. No imputation is planned for missing data and, unless unexpectedly high levels of missingness are observed, data will be assumed to be missing at random and missing data points will be excluded from the analysis. Available data for the primary outcome will be a requirement for all 3 patients at each dosing level before proceeding with the next dose. In keeping with methodologic guidelines for dose-finding studies, inferential analyses will not be performed and will focus instead on a non-frequentist confidence interval estimation approach.

### **Data monitoring**

Data will be reviewed after each dose by a data safety monitoring board (DSMB), who will confirm it is safe to escalate to the dose proposed using the Bayesian dose response model. The DSMB will be comprised of two emergency physicians and will be independent from the sponsor and reporting structure.

#### **METHODS: MONITORING**

#### Harms

### **Study Assessment and Procedures Assessment of Safety**

The onset of sedation, duration of sedation, maladaptive behaviors due to sedation, nasal irritation, vital signs are also important measures used to assess safety.

Onset of sedation: This will be defined as the time interval from administration of the first pair of IN sprays to the time when a PSSS score of 2 or 3 is achieved, whether or not all of the intervention has been administered. This will be ascertained by the outcome assessors.

<u>Duration of sedation</u>: This will be defined as the duration of time between the first PSSS score of 2 or 3 to the last PSSS score of 2 or 3 post-laceration repair. This will be ascertained by the outcome assessors.

<u>Maladaptive behaviors due to sedation</u>: This will be assessed by the research associate using the Post-Hospital Behavior Questionnaire (PBHQ) administered by phone or email survey 24 to 48 hours following discharge. This will be done in order to screen for any delayed behavioral adverse effects. This information will be recorded using REDCap (Dose Finding Study PHBQ form).

<u>Nasal irritation</u>: The research assistant will ask participants age  $\geq 4$  years using the Faces Pain Scale – Revised (FPS-R) to rate their nasal irritation related to the IN sprays. Nasal irritation has not been described with IN dexmedetomidine but is theoretically possible and needs to be identified in order to provide appropriate anticipatory guidance.

<u>Vital Signs</u>: Heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP) and oxygen saturation (SpaO2), respiratory rate (RR) will be recorded at baseline and every 5 minutes until 60 minutes after last pair of sprays is administered. Data will be collected using REDCap (Vital signs CRF form).

Adverse events (AEs): The research associate will be trained on the recognition and definition of all expected and unexpected AEs. AEs are document medical events that occur to a participant/subject once enrolled in a study. AEs are the construct through which the safety of an intervention is recorded and assessed during the study period.

Data will be collected using REDCap (Dose finding Study AE form). The form includes the definitions and AE descriptions that could be related to sedation. Uncertainty regarding the presence of AEs will be clarified with the sedating physician (if it occurs while participant is in the paediatric emergency department) and with PI for all AE cases reported. All AEs will be recorded.

### **Monitoring of Adverse Events During Sedation**

In two systematic reviews (11, 13) of intranasal dexmedetomidine in children (29 trials, 3134 participants), adverse cardiorespiratory events requiring intervention have not been described. This is in contrast to the use of IV dexmedetomidine and may be explained by the reduced bioavailability of the intranasal route (median 65%). However, to monitor the presence of serious adverse effects, several measures will be in place. Commencing immediately prior to administration of the intervention and continuing until the participant is awake, all participants will receive continuous cardiorespiratory monitoring. In accordance with our institutional policies

and recommendations from the American College of Emergency Physicians' Guidelines, this consists of

- 1. Five-lead continuous ECG to assess for the presence of bradycardia, dysrhythmias, and early changes suggestive of hypokalemia (< 3 mEq/L) (flattened or inverted T waves progressing to QT prolongation, ST depression, and U waves). If suggestive ECG changes are present, the participant will have a stat capillary puncture to measure the serum potassium.
- 2. Oxygen saturation to assess for the presence of desaturation
- 3. Blood pressure assessments using a Dynamap every 5 minutes to assess for the presence of hypotension or hypertension

A staff anesthetist is in house 24-7 in our institution. In the event that an adverse electrolyte or cardiopulmonary event is identified, the appropriate resuscitative measures will be provided based on the opinion and direction of the treating paediatric emergency physician. In our institution, resuscitative measures in the emergency department fall under the responsibility of the treating paediatric emergency physician. In the event of clinically significant hypokalemia, this may include but is not restricted to oral potassium chloride. In the event of clinically significant hypotension or bradycardia, this may include but is not restricted to reverse Trendelenberg positioning, placement of an intravenous line and administration of crystalloid fluids, and other measures consistent with the Paediatric Advanced Life Support algorithm.

### **Serious Adverse Event and Unexpected Drug Reactions**

A **Serious Adverse Event (SAE)** will be defined as - any adverse occurrence of a clinical trial subject who is administered a drug at any dose, or placebo that may or may not be caused by the administration of the drug or placebo that results in:

- 1. Hospitalization due to a sedation related event
- 2. Prolongation of existing hospitalization
- 3. Congenital malformation or birth defect
- 4. Persistent or significant disability or incapacity
- 5. An outcome that is life-threatening
- 6. Death

Important medical events that may not result in death, be life-threatening, substantially disrupt one's ability to conduct normal life functions or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

All serious, unexpected AEs and drug reactions will be reported to Health Canada by the Qualified Principal Investigator within 15 calendar days after the Qualified Principal Investigator becomes aware of the event. For death or life-threatening events, this report must be done within 7 calendar days after the Qualified Principal Investigator becomes aware of the event. In the latter

case, a follow-up report must be filed within 8 calendar days. All AEs will also be submitted, in accordance with the DSMB safety monitoring plan to the independent DSMB assigned to this study.

All serious adverse events (SAEs) will be followed until satisfactory resolution or until the PI deems the event to be chronic or the participant is stable. The Qualified Principal Investigator will also, within 8 days after having informed Health Canada of the adverse drug reaction, submit as complete as possible, a report which includes an assessment of the importance and implication of any findings.

A completed Adverse Drug Reaction (ADR) Expedited Reporting Summary Form should be attached to the front of the completed ADR report (suggested ADR report format: Suspect Adverse Reaction Report - CIOMS form of the Council for International Organizations of Medical Sciences (CIOMS)). Please find the form attached as Appendix C. **Adverse Events Reporting** 

All adverse events (AEs) will be reported to the Research Ethics Board in accordance with site's AE reporting guidelines. The PI will assess each AE in terms of its expectedness and relationship to the study drug. Information to be collected will include an event description, date of onset, clinician's assessment of severity, relationship to study intervention (assessed only by those with the training and authority to make a diagnosis), and date of resolution/stabilization of the event and event outcome (resolved/recovered, recovered with sequalae, not recovered/not resolved, death, or unknown).

### **Study Discontinuation and Closure**

This study may be temporarily suspended or prematurely terminated if there is sufficient reasonable cause based on the findings of the DSMB of safety issues. The latter include determination by the DSMB of significant adverse events that pose an unacceptable risk to participants such as complications due to treatment or related adverse events at rates above expected. Serious adverse events as defined by the Quebec Guidelines (16) on paediatric procedural sedation will be reported as per Good Clinical Practices. Data will be reviewed by the two-member DSMB prior to each planned dose increase. The two members will need to unanimously agree that it is safe to increase the dose. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party (DSMB) to study participants, funding agency (if applicable), the Sponsor, responsible REB and Health Canada. The Study participants will be contacted by Qualified Principal Investigator, as applicable, and be informed of changes to study visit schedule (if applicable). The study may resume once concerns about safety, protocol compliance, and data quality are addressed, and satisfy the Sponsor, REB and/or Health Canada.

### Withdrawal / Discontinuation Criteria

Participants are free to withdraw from participation in the study at any time upon request. However, data accrued from the participant to the time of withdrawal will be retained by the investigators for analysis. Example, if participant decided to withdraw the study before receiving the intranasal sprays. All data up to the point participant requested to be withdrawn will be kept. An investigator may discontinue or withdraw a participant from the study for the following reasons:

- 1. If any clinical adverse event (AE), laboratory abnormality, or other medical condition or situation occurs such that continued participation in the study would be detrimental to the health of the participant.
- 2. If the participant is found to meet exclusion criteria (either newly developed or not previously recognized) that precludes further study participation.

The reason for participant discontinuation or withdrawal from the study will be recorded on the Dose Finding Study Case Report Form (CRF- End of Study Form). For the purposes of this trial, a protocol violation will be defined as *any accidental or unintentional change or non-compliance with the REB approved protocol which increases or decreases benefit, affects the subject's rights, safety or welfare or the integrity of the study.* In the event that a participant is found to meet exclusion criteria (either newly developed or not previously recognized), this constitutes a protocol violation and the protocol will be discontinued. However, the participant will be followed for the study period for AEs. A protocol violation report must be completed as per local REB requirements and notification should be sent to the local REB (Western University - Research ethics board) by email. A note to file signed by the site PI should be completed and if any clinical adverse event (AE) occurs, an AE should also be completed and signed by PI and research staff. A copy of all documents must be sent to the local REB.

Follow up for participants withdrawn from investigational product: All participants who receive the interventional drug, including those who withdrawn, will be asked to remain in the emergency department until they are fully recovered from sedation as per the treating physician. Participants who are withdrawn after receiving interventional product will be contacted approximately 24 to 48 hours after discharge by a research associate via telephone. These participants will be asked an open-ended question such as: do you have any health concern since you were discharged from paediatric emergency department? If they return to the emergency department within 24 hours, the participant's medical record will be scrutinized by the research associate for adverse events as defined by the Quebec Guidelines (16) on paediatric procedural sedation.

Caregivers and participants will be advised at discharge and during the follow-up phone call that if they (or their child as applicable) experience adverse effects that they believe require a hospital visit, it is important that they make every effort to return to the hospital where procedure was performed. If they need immediate treatment and are unable to return to the hospital, they should proceed to the nearest emergency as soon as possible

### **Quality Assurance and Quality Control**

Quality control (QC) procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated to the site(s) for clarification/resolution.

Following written Standard Operating Procedures (SOPs), the monitors will verify that the clinical trial is conducted and data are generated, documented (recorded), and reported in compliance with the protocol, International Conference on Harmonisation Good Clinical Practice (ICH GCP), and applicable regulatory requirements.

The investigational site will provide direct access to all trial-related source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

All individuals from the research team such as site Investigator, site coordinators, and other research personnel will be required to complete the Tri-Council Policy Tutorial: Ethical Conduct for Research Involving Humans, the Good Clinical Practices course, and the division 5 Health Canada module. Completion will be documented prior to implementation of the study. Privacy and confidentiality policy and procedure will also be reviewed at the study recruitment training session for all study personnel.

### Auditing

The investigational site will provide direct access to all trial-related source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

### ETHICS AND DISSEMINATION

### **Statement of Compliance**

The trial will be conducted in accordance with Good Clinical Practice (GCP) as described in Health Canada's section C.05.010/Division 5 of the Food and Drugs Regulations, International Conference on Harmonization-Good Clinical Practice (ICH-GCP E6 R2), Tri-Counsel Policy Statement (TCPS2, 2014); applicable federal, provincial and local regulatory and legislative requirements. The Qualified and Participating Site Investigator(s) will assure that no deviation from, or changes to the protocol will take place without prior documented authorization (no objection letter - NOL) from Health Canada (Therapeutic Products Directorate) and documented approval from a duly constituted Research Ethics Board (REB), except where necessary to eliminate an immediate hazard(s) to the trial participants. All personnel involved in the conduct of this study have completed Human Subjects Protection and ICH-GCP Training.

### Research ethics approval

The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the REB for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled.

### **Protocol amendments**

Any amendment to the protocol will require review and approval by the REB before the changes are implemented to the study as well as authorization form Health Canada. All changes to the consent form will be REB approved; a determination will be made regarding whether a new consent needs to be obtained from participants who provided consent, using a previously approved consent form

### **Consent or assent**

If a patient is eligible, the Research Assistant will obtain informed consent and assent (when applicable).

### **Confidentiality**

Please refer to the data management section. All identifying participant information will be kept confidential in accordance with our REB requirements. The REDCap project will contain no identifying information.

### **Declaration of interests**

None

### Access to data

All electronic records and data sets will be encrypted and password protected with access only permitted by the PI, site coordinator(s), and research team members. The investigational site will provide direct access to all trial-related source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities

### Ancillary and post-trial care

Post-sedation care and monitoring will be in accordance with local institutional policies for sedated patients. Discharge instructions appropriate to laceration repair will be provided.

### **Dissemination policy**

Trial results in the form of an abstract will be presented at local research days and national scientific meetings. The manuscript will be submitted to a peer reviewed medical journal. Results will be disseminated informally to the study team and health care personnel at the participating site. There are no plans for dissemination of results directly to participants.

### References

- 1. Services USDoHaH. Centers for Disease Control and Prevention. National Survey of Ambulatory Surgery. 2015 [Available from: <a href="https://www.cdc.gov/nchs/nsas/nsas\_products.htm">https://www.cdc.gov/nchs/nsas/nsas\_products.htm</a>.
- 2. O'Donnell M WJ. Children's Emergency Department Services: Setting the Stage for Tiers Development Vancouver, BC.2016 [Available from: https://www.childhealthindicatorsbc.ca/sites/default/files/16%2010%2001%20ED%20Tiers%20S

https://www.childhealthindicatorsbc.ca/sites/default/files/16%2010%2001%20ED%20Tiers%20Setting%20the%20Stage 1.pdf.

- 3. Neville DNW, Hayes KR, Ivan Y, McDowell ER, RD P. Double-blind randomized controlled trial of intranasal dexmedetomidine versus intranasal midazolam as anxiolysis prior to pediatric laceration repair in the emergency department. Acad Emerg Med. 2016;23:910-7.
- 4. Taddio A, McGrath P, A. F. Effects of early pain experience: The human literature. Progress in Pain Research and Management. 1999;13:57-74.
- 5. Coté CJ, Wilson S, American Academy of Pediatrics, Dentistry AAoP. Guidelines for monitoring and management of pediatric patients before, during, and after sedation for diagnostic and therapeutic procedures: update 2016,. Pediatrics. 2016;138(1):e1-e31.
- 6. Miller JL CA, Thomas A, Couloures K, Johnson PN. Sedation and analgesia using medications delivered via the extravascular route in children undergoing laceration repair. J Pediatr Pharmacol Ther. 2018;23:72-83.
- 7. Conway A, Rolley J, JR S. Midazolam for sedation before procedures. Cochrane Database Syst Rev. 2016;5:CD009491.
- 8. Kogan A, Katz J, Efrat R, al. e. Premedication with midazolam in young children: a comparison of four routes of administration. Paediatr Anaesth. 2002;12:685-9.
- 9. Fantacci C, Fabrizio GC, Ferrara P, Franceschi F, A C. Intranasal drug administration for procedural sedation in children admitted to pediatric emergency room. Eur Rev Med Pharmacol Sci. 2018;22:217-22.
- 10. ter Bruggen FFJA, Eralp I, Jansen CK, Stronks DL, FJPM H. Efficacy of dexmedetomidine as a sole sedative agent in small diagnostic and therapeutic procedures: a systematic review. Pain Pract. 2017;17(6):829-40.
- 11. Kim HJ, Shin WJ, Park S, Ahn HS, JH O. The sedative effects of the intranasal administration of dexmedetomidine in children undergoing surgeries compared to other sedation methods: A systematic review and meta-analysis. J Clin Anesth. 2017;38:33-9.
- 12. Hayden JC, Breatnach C, Doherty DR, Healy M, Howlett MM, Gallagher PJ, et al. Efficacy of  $\alpha$ 2-agonists for sedation in pediatric critical care: a systematic review. Pediatr Crit Care Med. 2016;17(2):e66-75.
- 13. Spohn J, Hendrikx S, Doyon-Trottier E, Sabhaney V, Ali S, Shah A, et al. Intranasal dexmedetomidine for procedural distress in children: a systematic review and meta-analysis. CJEM. 2019;21(Suppl 1):S30.
- 14. Cravero JP AN, Sriswasdi P, Tsze DS, Zurakowski D, Sinnott S. Validation of the Pediatric Sedation State Scale. Pediatrics. 2017;139(5):e20162897.

- 15. O'Quigley H, Pepe M, Fisher L. Continual reassessment method: a practical design for phase 1 clinical trials in cancer. Biometrics. 1990;46(1):33-48.
- 16. Berry DA, Berry SM, Carlin BP, Lee JJ, Muller P. Bayesian Adaptive Methods for Clinical Trials. CRC Press LLC; 2010.
- 17. Yuen VM, Hui TW, Irwin MG, Yao TJ, Wong GL, MK Y. Optimal timing for the administration of intranasal dexmedetomidine for premedication in children. Anaesth. 2010;65(9):922-9.
- 18. Cheung YK. Sample size formulae for the Bayesian continual reassessment method. Clin Trials. 2013;10(6):852-61.
- 19. Bhatt M, Kennedy RM, Osmond MH, al. e, Network. CPoSRoPERCatPECAR. Consensus-based recommendations for standardizing terminology and reporting adverse events for emergency department procedural sedation and analgesia in children. Ann Emerg Med. 2009;53(4):426-35.e4.

### **APPENDICES**

### Appendix A

#### OFFICIAL JOURNAL OF THE AMERICAN ACADEMY OF PEDIATRICS

### PEDIATRICS<sup>®</sup>

### Intranasal dexmedetomidine for procedural distress in children: a systematic review

| Journal: | Pediatrics |
|---|---|
| Manuscript ID | 2019-1623.R2 |
| Article Type: | Review Article |
| Date Submitted by the<br>Author: | n/a |
| Complete List of Authors: | Poonai, Naveen; Western University Schulich School of Medicine and Dentistry, Paediatrics, Internal Medicine, Epidemiology & Biostatistics Spohn, Joseph; Western University Schulich School of Medicine and Dentistry, Paediatrics Vandermeer, Ben; University of Alberta, Pediatrics Ali, Samina; University of Alberta, Pediatrics Bhatt, Maala; Children's Hospital of Eastern Ontario, Pediatrics Hendrikx, Shawn; Western University Schulich School of Medicine and Dentistry, Paediatrics Trottier, Evelyne; Université de Montréal, CHU Sainte-Justine, Pediatrics Emergency Sabhaney, Vikram; The University of British Columbia, Paediatrics Shah, Amit; Western University Schulich School of Medicine and Dentistry, Internal Medicine Joubert, Gary; Children's Hospital, Emergency Medicine Hartling, Lisa; University of Alberta, Pediatrics |
| Keyword/Topic: | Anesthesiology/Pain Medicine |
| | <b>9</b> , |

SCHOLARONE™ Manuscripts

1 Title 2 Intranasal dexmedetomidine for procedural distress in children: a systematic review 3 Authors and Affiliations 5 Naveen Poonai MDa,b,c, Joseph Spohn MScb, Ben Vandermeer MScd, Samina Ali MDCMe,f, 6 Maala Bhatt MDg, Shawn Hendrikx MLISa, Evelyne D.Trottier MDCMh, Vikram Sabhaney 7 MDi, Amit Shah MDb, Gary Joubert MDa,b, Lisa Hartling PhDd 8 9 <sup>a</sup>Department of Pediatrics, Schulich School of Medicine and Dentistry, London, Canada <sup>b</sup>Division of Emergency Medicine, Western University, London, Canada 10 Children's Health Research Institute, London Health Sciences Centre, London, Canada 11 12 dAlberta Research Centre for Health Evidence (ARCHE), Department of Pediatrics, University 13 of Alberta, Edmonton, Canada Department of Pediatrics, Faculty of Medicine & Dentistry, University of Alberta, Edmonton, 14 15 Canada 16 <sup>f</sup>Women and Children's Health Research Institute, University of Alberta, Edmonton, Canada 17 EDepartment of Pediatrics, Children's Hospital of Eastern Ontario, Ottawa, Canada <sup>h</sup>Centre Hospitalier Universitaire Sainte-Justine, Université de Montréal, Canada 18 <sup>i</sup>BC Children's, University of British Columbia, Vancouver, Canada 19 20 21 Corresponding Author Dr. N. Poonai 22 Research Director, Division of Pediatric Emergency Medicine, Children's Hospital, London 23 Health Sciences Centre, London, Ontario 24 25 Associate Professor, Paediatrics and Internal Medicine, Schulich School of Medicine & 26 Dentistry, London, Ontario 27 800 Commissioners Road East, London, Ontario, Canada, N6A 2V5 Email: naveen.poonai@lhsc.on.ca 28 29 Phone: 519 685 8500 extension 52011 Fax: 519 667 6769 30 31 32 Short Title: Intranasal dexmedetomidine for procedural distress 33 34 Financial Disclosure: The authors have no financial relationships relevant to this article to 35 disclose 36 37 Funding Source: None 38 39 Conflict of Interest Statement: Potential Conflicts of Interest: The authors have no conflicts of 40 interest relevant to this article to disclose 41 42 Prospero Registry Number: CRD 42018102858 43 44 Abbreviations: 45 ABR auditory brainstem response CI confidence interval 46

| 47 | CT computed tomography |
|---|---|
| 48 | FLACC Faces Legs Activity Cry Consolability |
| 49 | GRADE Grading of Recommendations Assessment, Development, and Evaluation |
| 50 | IN intranasal |
| 51 | IND intranasal dexmedetomidine |
| 52 | IQR interquartile range |
| 53 | MAD mucosal atomizer device |
| 54 | IV intravenous |
| 55 | MRI magnetic resonance imaging |
| 56 | OR odds ratio |
| 57 | TTE transthoracic echocardiography |
| 58 | VEPs visually evoked potentials |
| 59 | |
| 60 | Table of Contents Summary: This systematic review of 19 trials (2137 participants) |
| 61<br>62 | summarized the effectiveness of intranasal dexmedetomidine for procedural distress in children. |
| 63 | What's Known on This Subject: Painful and distressing procedures are commonly performed |
| 64 | in children. Oral and intranasal midazolam, the most commonly used anxiolytics have limited |
| 65 | evidence of benefit. Intranasal dexmedetomidine is a relatively new agent but its study has been |
| 66 | limited by small sample sizes. |
| 67 | |
| 68 | What This Study Adds: Intranasal dexmedetomidine may provide more effective sedation than |
| 69 | chloral hydrate or midazolam. Limited data exist for minor, painful procedures such as laceration |
| 70 | repair or lumbar puncture. The benefits of administration must be weighed against the potential |
| 71 | for adverse cardiovascular effects. |
| 72 | |
| 73 | |
| 74 | |
| 75 | |
| 13 | |
| 76 | |
| 70 | |
| 77 | |
| , , | |
| 78 | |
| 79 | |
| 80 | |
| 81 | |
| 82 | |

| 83 | Contributor's Statement |
|---|---|
| 84<br>85<br>86<br>87<br>88<br>89<br>90<br>91<br>92<br>93 | Drs. Poonai, Ali, Hartling and Mr. Spohn conceptualized and designed the study, drafted the initial manuscript, and reviewed and revised the manuscript. Mr. Hendrikx conducted the literature search, and reviewed and revised the manuscript. Mr. Spohn designed the data collection instruments and collected data and reviewed and revised the manuscript. Mr. Vandermeer carried out the initial analyses and reviewed and revised the manuscript. Drs. Joubert, D.Trottier, Shah, Sabhaney, and Bhatt critically reviewed the manuscript for important intellectual content. All authors approved the final manuscript as submitted and agree to be accountable for all aspects of the work. |
| 95 | |
| 96 | |
| 97 | |
| 98 | |
| 99 | |
| 100 | |
| 101 | |
| 102 | |
| 103 | |
| 104 | |
| 105 | |
| 106 | |
| 107 | |
| 108 | |
| 109 | |
| 110 | |

| 111 | ABSTRACT |
|---|---|
| 112<br>113 | Context: Intranasal dexmedetomidine (IND) is an emerging agent for procedural distress in children. |
| 114 | |
| 115 | Objective: To explore the effectiveness of IND for procedural distress in children. |
| 116 | D. C. W. C. A. C. C. A. C. |
| 117 | Data Sources: We performed electronic searches of MEDLINE (1946-2019), EMBASE (1980- |
| 118 | 2019), Google Scholar (2019), CINAHL (1981-2019), and Cochrane Central Register. |
| 119<br>120 | Study Selection: We included randomized trials of IND for procedures in children. |
| 121 | Study Selection: We included fandomized thats of IND for procedures in children. |
| 122 | Data Extraction: Data extraction was performed in duplicate. Methodological quality and |
| 123 | quality of evidence were evaluated using the Cochrane Collaboration's Risk of Bias tool and the |
| 124 | Grading of Recommendations Assessment, Development, and Evaluation system, respectively. |
| 125 | The primary outcome was the proportion of participants with adequate sedation. |
| 126 | The primary concerns was the proportion of participants with medical securion. |
| 127 | Results: Among 19 trials (n=2137), IND was superior to oral chloral hydrate (3 trials), oral |
| 128 | midazolam (one trial), intranasal midazolam (one trial), and oral dexmedetomidine (one trial). |
| 129 | IND was equivalent to oral chloral hydrate (two trials), intranasal midazolam (two trials), and |
| 130 | intranasal ketamine (three trials). IND was inferior to oral ketamine and a combination IND plus |
| 131 | oral ketamine (one trial). Higher doses of IND were superior to lower doses (four trials). Adverse |
| 132 | effects were reported in 67/727 (9.2%) participants in the IND versus 98/591 (16.6%) in the |
| 133 | comparator group. There were no reports of adverse events requiring resuscitative measures. |
| 134 | |
| 135 | Limitations: Adequacy of sedation was subjective; possibly leading to biased outcome |
| 136 | reporting. |
| 137 | |
| 138 | Conclusions: Given the methodological limitations of included trials, IND is likely more |
| 139 | effective at sedating children compared to oral chloral hydrate and oral midazolam. However, |
| 140 | this must be weighed against the potential for adverse cardiovascular effects. |
| 141 | |
| 142 | |
| 143 | |
| 144 | |
| 145 | |
| 146 | |
| 147 | |
| 148 | |

### INTRODUCTION

149

150

151

152

153

154

155

156

157

158

159

160

161

162

163

164

165

166

167

168

169

170

171

In hospital, painful and distressing procedures including laceration repair, lumbar puncture (1), intravenous (IV) insertion (2-6), and venipuncture (6, 7) are common. However, administration of analgesia is inconsistent for painful procedures and procedural distress is poorly managed (2-6). A Canadian survey of over 3000 hospitalized children found that they received more than six painful procedures per day, and less than one third of them received analgesia (8). Such procedures result not only in the reported pain, but also in closely-linked procedural distress, which often requires a different approach than simply analgesia. Further, other non-painful diagnostic procedures, such as CT and magnetic resonance imaging (MRI), require a child to lie motionless which can be anxiety-provoking across the age spectrum, and often requires some level of sedation for younger patients. To address these issues of sedation and anxiolysis, intranasal (IN) therapies for procedural distress can be non-invasively administered (9) and require less procedural skill than IV insertion (10). Currently, midazolam is the most commonly used anxiolytic in children because of its rapid onset of action and amnestic properties (11). However, when used via the IN route, it has an unpleasant taste, can be irritating to the nasal mucosa (12, 13), and has adverse effects (11, 14), underscoring the need for appropriate monitoring. Furthermore, two Cochrane reviews have differing conclusions regarding midazolam's effectiveness for children's procedures (11, 14), suggesting that additional evidence for alternative agents is needed. Dexmedetomidine is a central α<sub>2</sub>-adrenergic receptor agonist with analgesic and anxiolytic properties and its use outside the intensive care and pre-anesthetic setting is gaining popularity (15). Three systematic reviews suggest dexmedetomidine, is effective for procedural

distress in children (15-17). However, they mainly reported effects by IV route and only one explored intranasal dexmedetomidine (IND), focusing on anesthetic premedication (16). To date, no large trial or review exists to guide the use of IND for procedural distress in children. With the emerging popularity of dexmedetomidine for procedural distress and a desire for less invasive approaches in children, a comprehensive review of IND is needed to guide its use. We sought to summarize the effectiveness of IND for children undergoing painful and distressing procedures.

#### PATIENTS AND METHODS

This review followed the Preferred Reporting Items for Systematic Reviews and Meta-Analysis guidelines (18) (Appendix 1).

#### Eligibility Criteria

We included all published and unpublished randomized trials comparing IND as monotherapy to any comparator for a procedure in children under 19 years and reported adequacy of sedation. Trials of both adults and children were included if the authors provided pediatric-specific data. We excluded sub-studies, crossover studies, abstracts with insufficient information, and studies of anesthetic premedication unless they involved a painful procedure.

The primary outcome was the proportion of participants deemed to be adequately sedated based on the investigators' opinion. Clinically, we believed this to be the most pragmatic, relevant, and feasible approach to describing relief of procedural distress. Methodologically, we believed this to be consistent way of overcoming differences in sedation scales. Secondary outcomes included need for additional sedation, onset and duration of sedation, length of stay, analgesia, adverse events, and acceptance of IN administration.

### Data Sources

195 A medical librarian (SH) developed the search strategy. We performed electronic 196 searches of MEDLINE (1946 - 2018), EMBASE (1980 - 2018), Scopus (2018), Web of Science 197 (2018), Google Scholar (2018), Cochrane Central Register (2018), and CINAHL (1981 to 2018). 198 The search was completed in January 2018 and repeated in February and July 2019 without 199 language restriction (Appendix 2). Our gray literature search was informed by the Canadian 200 Agency for Drugs and Technologies in Health checklist (19). We checked reference lists of 201 included trials and systematic reviews. We contacted corresponding authors when data on the 202 primary outcome was missing. 203 Study Selection and Data Extraction 204 Two authors (NP, JS) independently screened titles, abstracts, and full-texts for inclusion. 205 Disagreements were resolved through discussion. The primary author entered the data into 206 Review Manager version 5.2.11 and GRADEpro version 3.6. 207 Risk of Bias in Individual Studies 208 Two authors (NP, JS) independently evaluated methodological rigor using the Cochrane 209 Collaboration's Risk of Bias tool (20) and outcome-specific ratings of the overall quality of 210 evidence using the Grading of Recommendations Assessment, Development, and Evaluation 211 (GRADE) system (21). 212 Summary Measures and Synthesis of Results 213 A priori we considered meta-analyses if there was homogeneity in procedures, dosing 214 regimen, and outcome measures. However, meta-analyses were not performed on any outcome 215 due to substantial heterogeneity. Instead, we conducted a descriptive analysis of each study's 216 design, population, and primary outcome. Based on the classification system of Tricco et al. (22), 217 we categorized the results of individual studies based on the outcome of adequate sedation as:

218 unfavorable (effect in favor of the comparator with p value  $\leq 0.05$ ); neutral (non-statistically 219 significant difference between interventions with p value > 0.05)); favorable (effect in favor of 220 the experimental agent, IND, with p value  $\leq 0.05$ ); indeterminate (unable to judge due to 221 conflicting and multiple primary outcomes). We used ranges to describe onset and duration of 222 sedation and length of stay. We used proportions to describe acceptance of IN administration. 223 Agreement between reviewers was described using raw agreement. 224 Risk of Bias Across Studies 225 Publication bias was assessed using a funnel plot. 226 Additional Analyses 227 We evaluated statistical heterogeneity using the  $I^2$  statistic. 228 RESULTS 229 Study Selection 230 Nineteen trials (n=2137) were included. Thirteen involved IND versus a non-IND 231 comparator. Six compared different doses of IND or methods of IND administration (Figure 1). 232 Study Characteristics 233 IND was studied for the following non-painful procedures: ophthalmic examination (3 234 trials) (23-25); transthoracic echocardiography (TTE) (2 trials) (26, 27); auditory brainstem 235 response (ABR) testing (2 trials) (28, 29); computed tomography (CT) (3 trials) (29-31), 236 magnetic resonance imaging (MRI) (2 trials) (32, 33); visually evoked potentials (VEPs) (1 trial) 237 (29) and was studied for the following painful procedures: IV insertion (6 trials) (31, 34-38), 238 laceration repair (1 trials) (39), and dental work (2 trials) (40, 41). All trials were published in 239 English in peer reviewed journals and included 2137 children (847/2093, 40.5% females), age 1 240 month to 14 years. Demographic statistics excluded Patel et al. (41) because these details were

241 not specified. IND was compared to oral dexmedetomidine (41), chloral hydrate (23, 26, 28, 30, 242 33), IND plus oral ketamine (37), IN or oral midazolam (31, 34, 39, 40), IN or oral ketamine (35-243 37, 40). Six trials compared different doses of IND (24, 25, 29, 32) or methods of IND 244 administration (27, 38) (Table 1). 245 Risk of Bias Within Studies 246 Most trials were judged as low risk of bias for random sequence generation, blinding, 247 incomplete outcome data, and selective reporting (Figure 2). For allocation concealment, most 248 trials were judged as unclear risk of bias. Li et al. was judged as high risk of bias for incomplete 249 outcome data because 14/67 participants receiving IND 1 mcg/kg withdrew post-randomization 250 with no outcome data reported (29). Surendar et al. reported vital signs instead of adverse effects 251 and was judged as unclear risk of bias (40). 252 Risk of Bias Across Studies 253 The overall quality of evidence based on the GRADE system was judged as high (length 254 of stay), moderate (need for additional sedation, duration of sedation, and adverse effects), or 255 low (adequacy of sedation, onset of sedation, and analgesia) (Figure 3). 256 Adequacy of Sedation 257 Adequacy of sedation was reported in 18 of 19 trials. A validated sedation instrument 258 was used in ten trials (25-27, 29-34, 36) and included the Observer's Assessment of 259 Alertness/Sedation, Modified Observer's Assessment of Alertness/Sedation Scale, Ramsay 260 Sedation Scale, and the University of Michigan Sedation Scale (Table 1). Seven trials used non-261 validated scales to measure sedation (24, 28, 35-37, 40, 41). Two trials did not report adequacy 262 of sedation but pain during IV insertion using the Faces Legs Activity Cry Consolability 263 (FLACC) scale (38) and anxiety during early stages of laceration repair using the Yale

| 264 | Preoperative Anxiety Scale (YPAS) (39). The proportion of participants with adequate sedation |
|---|---|
| 265 | was 33/41 (80.4%) for IND plus oral ketamine, 1086/1362 (79.7%) for IND, 241/318 (75.7%) |
| 266 | for chloral hydrate, 28/41 (68.3%) for oral ketamine, 59/102 (57.8%) for intranasal ketamine, |
| 267 | 30/69 (43.4%) for intranasal midazolam, 7/29 (24.1%) for oral midazolam, and 0/22 (0%) for |
| 268 | oral dexmedetomidine. IND was deemed "favorable" versus chloral hydrate in three trials (23, |
| 269 | 28, 33), oral midazolam in one trial (31), intranasal midazolam in one trial (34), and oral |
| 270 | dexmedetomidine in one trial (41). IND was deemed "neutral" versus chloral hydrate in two |
| 271 | trials (26, 30), intranasal midazolam in two trials (39, 40), and intranasal ketamine in three trials |
| 272 | (35, 36, 40). IND was deemed "unfavorable" versus oral ketamine and a combination IND plus |
| 273 | oral ketamine in one trial (37). |
| 274 | Adequacy of Sedation for Painful and Non-Painful Procedures |
| 275 | For painful procedures (31, 34-41), IND provided adequate sedation to 145/237 (61.2%) |
| 276 | versus 151/321 (47.1%) participants among comparators. For non-painful procedures (23-33), |
| 277 | IND provided adequate sedation to 862/1025 (84.1%) versus 250/347 (72.0%) participants |
| 278 | among comparators. Limiting the comparison of painful versus non-painful procedures to trials |
| 279 | using validated instruments, IND versus comparators provided adequate sedation to 24/30 (80%) |
| 280 | versus 16/30 (53.3%) participants (painful), and 874/1021 (85.6%) versus 214/277 (77.3%) |
| 281 | participants (non-painful), respectively. |
| 282 | Differing Doses of IND and Routes of Nasal Administration |
| 283 | Six trials compared different doses or routes of IND administration. Gan et al. found that |
| 284 | 2 mcg/kg provided adequate sedation to significantly more participants undergoing |
| 285 | ophthalmologic examination than 1 mcg/kg (28/30, 93% versus 20/30, 67%, respectively; |
| 286 | p=0.02) (24). Chen et al. found that 2 and 3 mcg/kg provided a similar degree of sedation for |

| 287 | ophthalmologic examination; successfully sedating 49/50 (98%) and 50/50 (100%) participants, |
|---|---|
| 288 | respectively (25). Tug et al. found IND 4 mcg/kg provided adequate sedation to significantly |
| 289 | more participants undergoing MRI than 3 mcg/kg (20/30, 66.7% versus 7/30, 23.3%, |
| 290 | respectively; p=0.003) (32). Li et al. found that higher doses of IND (1 versus 1.5 versus 2 |
| 291 | mcg/kg) provided adequate sedation to increasingly more participants undergoing CT scan, ABR |
| 292 | testing, or VEPs [56/67 (83.6%), 66/74 (89.2%), and 51/53 (96.2%), respectively; p=0.03] (29). |
| 293 | Li et al. found no differences in adequate sedation for IND 3 mcg/kg by mucosal atomizer device |
| 294 | (MAD) or nasal drops [113/137 (82.5%) versus 120/142 (84.5%), respectively; p=0.57] (27). Xie |
| 295 | et al. found that the median (IQR) FLACC scores were significantly better with IND 2 mcg/kg |
| 296 | via an MAD versus nasal drops for IV insertion [1 (0.4) versus 3 (4); p=0.02, respectively] (38). |
| 297 | Need for Additional Sedation |
| 298 | Five trials reported on the need for additional sedation (26, 28, 31, 36, 39). Additional |
| 299 | sedation was provided to significantly fewer participants in the IND (22/223, 9.9%) versus |
| 300 | comparator groups (47/167, 28.1%). |
| 301 | Onset of Sedation |
| 302 | Onset of sedation was reported in 11 trials (23, 25, 26, 28, 30, 33, 34, 36, 37, 40, 41) and |
| 303 | ranged from 7-31 minutes for IND and 7-44.2 minutes for comparators. Onset of sedation varied |
| 304 | by dose of IND: 1 mcg/kg (14.3-19 minutes) (24, 29, 33, 34, 40), 1.5 mcg/kg (18.1-20 minutes) |
| 305 | (29, 40), 2 mcg/kg (8.8-25 minutes)(23-26, 29, 33, 38, 41), 2.5 mcg/kg (7-20.6 minutes) (37, 41), |
| 306 | 3 mcg/kg (13-31 minutes) (25-28, 30, 32, 36), and 4 mcg/kg (30 minutes) (32). |
| 307 | Duration of Sedation |
| 308 | Duration of sedation was reported insix trials (23, 25, 26, 33, 36, 40) and ranged from 41- |
| 309 | 91.5 minutes for IND and 77-85.9 minutes for comparators. |

| 310 | Length of Stay |
|---|---|
| 311 | Length of stay was reported in four trials (23, 24, 26, 39) and ranged from 76.8-156 |
| 312 | minutes for IND and 95-144 minutes for comparators. |
| 313 | Analgesia |
| 314 | Analgesia was reported using the FLACC scale by Surendar et al. (40) in children |
| 315 | undergoing dental procedures and Xie et al. (38) in children undergoing IV insertion. The |
| 316 | FLACC scale is scored from 0 to 10, with higher scores denoting greater pain (42). Using a |
| 317 | pairwise comparison, Surendar et al. reported mean (SD) FLACC scores for IND 1 mcg/kg [3.8 |
| 318 | (0.8)], 1.5 mcg/kg [3.7 (0.9)], and IN ketamine 5 mg/kg [3.5 (0.7)] were significantly lower than |
| 319 | IN midazolam 0.2 mg/kg [5.6 (1.1)] (p value not reported) (40). Xie et al. reported a lower |
| 320 | median (IQR) FLACC score for IND 2 mcg/kg by MAD [1 (3.5)] versus nasal drops [3 (4)] |
| 321 | (p=0.02) (38). |
| 322 | Adverse Events |
| 323 | Adverse events were reported in all trials except Surendar et al. (40). Across the |
| 324 | remaining 18 trials, the most common adverse events of IND, IND plus another sedative, or non |
| 325 | IND comparator were bradycardia [32/1484 (2.2%), 0/41 (0%), and 6/595 (1%), respectively], |
| 326 | $hypotension \ [18/1484\ (1.2\%),\ 0/41(0\%),\ and\ 9/595\ (1.5\%),\ respectively],\ oxygen\ desaturation$ |
| 327 | [7/1484 (0.5%), 0/41 (0%), and 12/595 (2%), respectively], and vomiting [6/1484 (0.4%), 3/41 |
| 328 | (7.3%), and 47/595 (7.9%), respectively]. No trials used objective criteria to define adverse |
| 329 | events. No trials reported the occurrence of upper airway obstruction, apnea, death, the delivery |
| 330 | of positive pressure ventilation, chest compressions, vasoactive medications, endotracheal |
| 331 | intubation, or neuromuscular blockade. |
| 332 | Acceptance of IN Administration |

333 Four trials reported acceptability of IN administration. Zhang et al. reported all 94 334 participants tolerated IND "without crying" (33). Xie et al. reported 25/49 (51%) versus 22/57 335 (38.6%) participants "calmly accepted" IND using an MAD versus drops, respectively (38). 336 Patel et al. reported acceptance of IND was "fair to excellent" in 16/22 (72.7%) of participants. 337 Surendar et al. reported IND and IN midazolam were "well accepted" by all 84 participants (40). 338 Agreement Between Reviewers 339 Two independent reviewers (NP, JS) agreed 102/114 (89.5%) times on risk of bias 340 assessments, 366/430 (85.1%) times on abstract screening and 74/79 (93.7%) times on full-text 341 screening. 342 Publication Bias 343 The funnel plot for adequacy of sedation showed some asymmetry (Appendix 3). 344 DISCUSSION 345 In this review, the overall quality of evidence for adequacy of sedation was "low". 346 Although our findings suggest that IND likely provides adequate sedation to a greater proportion 347 of children than conventional sedatives (oral midazolam and chloral hydrate), trial results could 348 not be pooled and larger and more methodologically rigorous trials are needed prior to 349 widespread implementation. Clinicians considering the use of IND to alleviate procedural 350 anxiety in children must weigh the benefit of superior sedation against the potential for adverse 351 cardiovascular effects, which require further rigorous study to fully assess the risk. 352 We chose to include trials that used midazolam and chloral hydrate as comparators 353 because they are widely used in clinical practice (43). In fact, chloral hydrate is recommended by 354 the National Institute for Health and Care Excellence (NICE) 2010 guideline for moderate 355 sedation for painless procedures in children (44). While chloral hydrate is no longer approved by

356

357

358

359

360

361

362

363

364

365

366

367

368

369

370

371

372

373

374

375

376

377

378

the United States Food and Drug Administration, it may still be used in other countries. IND provided adequate sedation in 79.7% of children, greater than that of chloral hydrate (75.7%), oral (24.1%) and intranasal midazolam (43.4%). This is consistent with a recent systematic review where IND was superior to oral benzodiazepines in children undergoing anesthetic premedication (16), as well as with another systematic review which found inconsistent evidence of procedural anxiolysis for IN midazolam (11), and with a trial of 300 children undergoing ABR. testing where IND sedated significantly more children than chloral hydrate (91% versus 78.5%, respectively) (45). IND may be a safer alternative to chloral hydrate given the latter's propensity to cause respiratory depression (46) and other major adverse effects such as bradycardia, hypotension, and oxygen desaturation (47). In response to evidence that general anesthetics and sedatives in young children may have adverse neurodevelopmental consequences, in 2016, the US Food issued a Drug Safety Communication mandating label changes for all anesthetic gases, and the IV agents propofol, ketamine, barbiturates, and benzodiazepines (48). Dexmedetomidine has been shown to be neuroprotective in animal studies (49) but little long-term data in humans exists. Although IND was reported to produce adequate sedation in more children than IN ketamine (79.7% versus 57.8%), IND was deemed "neutral" versus IN ketamine in all trials that compared the two agents (35, 36, 40). Each trial was small and may not have been sufficiently powered to detect differences in sedation. IND however, may be more suitable than IN ketamine for uncooperative children because fewer IN sprays are required. At 100 mcg/mL, an IND dose of 4 mcg/kg in a 25 kg child would only require two 0.5 mL sprays. Interestingly, in a single study of children undergoing IV insertion, IND was deemed "unfavorable" compared to a combination of IND and oral ketamine, with the latter producing adequate sedation in 80.4% of children (37). The sedative effects of dexmedetomidine may have complemented the well-known

379 analgesic effects of IN ketamine (50, 51) and future studies should explore the sedative potential 380 of this novel therapeutic combination. 381 The most effective non-invasive approach to providing dexmedetomidine appeared to be 382 the IN route. Although informed by only one trial, oral dexmedetomidine was unsuccessful in all 383 cases (41). Oral absorption of dexmedetomidine is possible (52) but its bioavailability is reduced 384 by first-pass metabolism (53). What remains unclear is whether IND administration using an 385 MAD is more efficacious than nasal drops. Li et al. found no difference among children 386 undergoing TTE, a relatively painless procedure (27). In contrast, Xie et al. found lower pain 387 scores during IV insertion using an MAD (38). Nasal drops may result in excess volume entering 388 the oropharynx and more difficult administration in uncooperative patients. Conversely, the 389 MAD takes advantage of the nasal cavity's large mucosal surface area and rich vascular supply 390 (13, 54, 55), resulting in a median bioavailability of 65% (53). 391 Insight into the analgesic potential of IND was limited to two trials that reported lower 392 FLACC scores with IND versus IN midazolam for dental procedures (40) and IND using an 393 MAD versus drops for IV insertion (38). Reduced opioid requirements have been reported with 394 IND in children post-adenotonsillectomy (56) and adults post-hip arthroplasty (57). IV 395 dexmedetomidine has also been shown to reduce opioid requirements in children undergoing 396 scoliosis repair (58) and cardiac surgery (59). However, the proportion of participants deemed as 397 being adequately sedated for painful versus non-painful procedures (61.2% versus 84.1%) 398 suggests that sedation using IND may be improved upon by the addition of a more potent 399 analgesic, perhaps one with sedative properties. Currently, IND as monotherapy is not indicated 400 for severely painful procedures and its analgesic potential appears to be realized in conjunction
401 with local anesthetics (60). Future studies should explore the analgesic potential of IND for 402 acutely painful procedures using rigorous methodology and optimal dosing. 403 The onset and duration of sedation are important considerations in a busy acute care 404 setting. We found wide ranges in onset and duration of IND (7-31 and 41-91.5 minutes, 405 respectively) and data did not support a dose effect. This may reflect heterogeneity in dosing or 406 definitions of sedation but are consistent with previous reports. Among healthy adult males, 407 Iirola et al. reported a median (range) peak plasma concentration at 38 (15-60) minutes and onset 408 of sedation of 30-45 minutes (53). In children, Yuen et al. reported a median (95% CI) onset and 409 duration of sedation of 25 (25 to 30) and 85 (55 to 100) minutes, respectively (61). These results 410 suggest that IND should be administered at least 30 minutes prior to an anxiety-provoking 411 procedure (53). The American Academy of Pediatrics has published guidelines outlining 412 monitoring requirements for children undergoing procedural sedation. Regardless of agent or 413 route of administration, all children should receive comprehensive monitoring for the duration of 414 sedation. This should include, but is not limited to, pulse oximetry and capnography (62). 415 Acceptance of IN administration was only assessed in four trials and not objectively. 416 However, there is good reason to believe that intolerance of nasal sprays is unlikely to preclude 417 IND administration because the drug is tasteless, odorless and painless (53, 54) and reportedly 418 "not noxious to the nasal mucosa" (53, 63), a notable difference from IN midazolam in which 419 discomfort is commonly reported (12, 13). 420 Adverse effects identified in our review such as bradycardia, hypotension, and 421 desaturation were reported across the dosing range and are likely to inform bedside monitoring 422 requirements. For the adverse cardiovascular effects we identified, no resuscitative maneuvers 423 were reported, suggesting they were self-resolving. This is consistent with two paediatric

424 systematic reviews that reported no respiratory compromise with either IND (16) or IV 425 dexmedetomidine (15). In addition, several pediatric studies found that IV dexmedetomidine was 426 associated with bradycardia without hemodynamic instability (15, 54, 58, 64, 65). Nevertheless, 427 it is difficult to know to what degree these occurrences compromised patient care. The most 428 prudent approach would be to limit the use of IND to children without cardiac conduction 429 anomalies, bradycardia, hypotension, or concomitant use of sympatholytic agents. Future studies 430 should define adverse events and corresponding interventions based on published guidelines 431 (66). 432 Limitations 433 Our review included a large number of small studies with some methodological 434 shortcomings, the most notable of which was subjective determination of adequacy of sedation. 435 The lack of a consistent and objective determination of this parameter may have led to biased 436 outcome reporting for this and other related outcomes such as onset and duration of sedation. 437 Due to heterogeneity in dosing and indications, it was difficult to appreciate differences in 438 adequate sedation among trials that used validated sedation instruments versus trials that did not. 439 However, based on the classification system outlined by the American College of Emergency 440 Physicians Clinical Policy, we believe that across trials, adequate sedation most closely 441 paralleled dissociative sedation, with the caveat that few trials determined the degree of 442 analgesia and no trials assessed amnesia (67). We found large heterogeneity across studies which 443 may be due to different comparators. The funnel plot showed some asymmetry, suggesting the 444 potential for publication or small study bias. As such, we downgraded our certainty of the 445 evidence for some outcomes.

https://mc.manuscriptcentral.com/pediatrics

446

Conclusions

447 Our findings suggest that IND is well-tolerated and may provide more effective sedation 448 than midazolam and chloral hydrate for distressing procedures in children. However, the quality 449 of evidence was "low" and larger, more methodologically rigorous trials are needed. The 450 available limited data for painful procedures (mostly IV insertion), suggests that while IND may 451 provide reasonable sedation, it may not provide adequate analgesia as monotherapy. As such, 452 more study is urgently required to understand the role of IND, perhaps in combination with a 453 more widely studied analgesic sedative for painful procedures. Transient cardiovascular adverse 454 effects, without reports of resuscitative intervention, were identified, and more rigorously 455 designed trials with standardized and objective reporting of adverse effects are needed to inform 456 the safe use of IND in children. 457 References 458 459 Ali S, Chambers AL, Johnson DW, Craig WR, Newton AS, Vandermeer B, et al. 1. 460 Paediatric pain management practice and policies across Alberta emergency departments. 461 Paediatrics & child health. 2014;19(4):190-4. Fradet C, McGrath PJ, Kay J, Adams S, Luke B. A prospective survey of reactions to 462 463 blood tests by children and adolescents. Pain. 1990;40(1):53-60. 464 Goodenough B, Thomas W, Champion GD, Perrott D, Taplin JE, von Baeyer CL, et al. 465 Unravelling age effects and sex differences in needle pain: ratings of sensory intensity and 466 unpleasantness of venipuncture pain by children and their parents. Pain. 1999;80(1):179-90. 467 Humphrey GB, Boon CM, van Linden van den Heuvell GF, van de Wiel HB. The 468 occurrence of high levels of acute behavioral distress in children and adolescents undergoing 469 routine venipunctures. Pediatrics. 1992;90(1 Pt 1):87-91. 470 Van Cleve L, Johnson L, Pothier P. Pain responses of hospitalized infants and children to 471 venipuncture and intravenous cannulation. Journal of Pediatric Nursing. 1996;11(3):161-8. 472 Friedrichsdorf SJ, Postier A, Eull D, Weidner C, Foster L, Gilbert M, et al. Pain 473 Outcomes in a US Children's Hospital: A Prospective Cross-Sectional Survey. Hospital 474 pediatrics. 2015;5(1):18-26. 475 Fein JA, Zempsky WT, Cravero JP, Medicine CoPEM, Section on A, Pain, et al. Relief 476 of pain and anxiety in pediatric patients in emergency medical systems. Pediatrics. 477 2012;130(5):e1391-405. 478 Stevens BJ, Abbott LK, Yamada J, Harrison D, Stinson J, Taddio A, et al. Epidemiology 479 and management of painful procedures in children in Canadian hospitals. CMAJ: Canadian 480 Medical Association journal = journal de l'Association medicale canadienne. 2011;183(7):E403-481 10.

- Del Pizzo J, Callahan JM. Intranasal Medications in Pediatric Emergency Medicine.
- 483 Pediatric Emergency Care. 2014;30(7):496-501.
- Murphy AP, Hughes M, McCoy S, Crispino G, Wakai A, O'Sullivan R. Intranasal
- 485 fentanyl for the prehospital management of acute pain in children. European Journal of
- 486 Emergency Medicine. 2016:1.
- Conway A, Rolley J, JR S. Midazolam for sedation before procedures. Cochrane
- 488 Database Syst Rev. 2016;5:CD009491.
- Kogan A, Katz J, Efrat R, al. e. Premedication with midazolam in young children: a
- 490 comparison of four routes of administration. Paediatr Anaesth. 2002;12:685-9.
- Fantacci C, Fabrizio GC, Ferrara P, Franceschi F, A C. Intranasal drug administration for
- 492 procedural sedation in children admitted
- 493 to pediatric emergency room. Eur Rev Med Pharmacol Sci. 2018;22:217-22.
- Ashley PF, Chaudhary M, L L-M. Sedation of children undergoing dental treatment.
- 495 Cochrane Database Syst Rev. 2018;12.
- 496 15. ter Bruggen FFJA, Eralp I, Jansen CK, Stronks DL, FJPM H. Efficacy of
- 497 dexmedetomidine as a sole sedative agent in small diagnostic and therapeutic
- 498 procedures: a systematic review. Pain Pract. 2017;17(6):829-40.
- 499 16. Kim HJ, Shin WJ, Park S, Ahn HS, JH O. The sedative effects of the intranasal
- 500 administration of dexmedetomidine in children undergoing surgeries compared to other sedation
- 501 methods: A systematic review and meta-analysis. J Clin Anesth. 2017;38:33-9.
- 502 17. Hayden JC, Breatnach C, Doherty DR, Healy M, Howlett MM, Gallagher PJ, et al.
- 503 Efficacy of α2-agonists for sedation in pediatric critical care: a systematic review. Pediatr Crit
- 504 Care Med. 2016;17(2):e66-75.
- Panic N, Leoncini E, de Belvis G, Ricciardi W, Boccia S. Evaluation of the Endorsement
- 506 of the Preferred Reporting Items for Systematic Reviews and Meta-Analysis (PRISMA)
- 507 Statement on the Quality of Published Systematic Review and Meta-Analyses. PLOS ONE.
- 508 2013;8(12):e83138.
- Canadian Agency for Drugs and Technologies in Health. Grey matters: a practical tool
- 510 for searching health-related grey literature 2018 [updated August 17, 2018]. Available from:
- 511 <a href="https://www.cadth.ca/resources/finding-evidence/grey-matters">https://www.cadth.ca/resources/finding-evidence/grey-matters</a>.
- 512 20. Julian PTH, Altman DG, Gøtzsche PC, Jüni P, Moher D, Oxman AD, et al. The Cochrane
- 513 Collaboration's tool for assessing risk of bias in randomised trials. BMJ: British Medical Journal.
- 514 2011;343(7829):889-93.
- Guyatt GH, Oxman AD, Vist GE, Kunz R, Falck-Ytter Y, Alonso-Coello P, et al.
- 516 GRADE: an emerging consensus on rating quality of evidence and strength of recommendations.
- 517 BMJ (Clinical research ed). 2008;336(7650):924-6.
- Tricco AC, Tetzlaff J, Pham B, Brehaut J, Moher D. Non-Cochrane vs. Cochrane reviews
- 519 were twice as likely to have positive conclusion statements: cross-sectional study. Journal of
- 520 Clinical Epidemiology. 2009;62(4):380-6.e1.
- Cao Q, Lin Y, Xie Z, Shen W, Chen Y, Gan X, et al. Comparison of sedation by
- 522 intranasal dexmedetomidine and oral chloral hydrate for pediatric ophthalmic examination.
- 523 Pediatr Anesth. 2017;27(629-36).
- 524 24. Gan X, Lin H, Chen J, Lin Z, Lin Y, W C. Rescue sedation with intranasal
- 525 dexmedetomidine for pediatric ophthalmic examination after chloral hydrate failure: a
- 526 randomized controlled trial. Clin Ther. 2016;38(6):1522–9.

Study: Intranasal dexmedetomidine for laceration repair in children: a dose finding study

Protocol: Dose Finding Study Version 3.5 – November 1, 2019

- 527 25. Chen C, You M, Li Z, Zhao Y, G C. Study of feasibility and safety of higher-dose
- 528 dexmedetomidine in special outpatient examination of pediatric ophthalmology. J
- 529 Ophthalmology. 2019.
- 530 26. Miller J, Xue B, Hossain M, Zhang M-Z, Loepke A, D K. Comparison of
- 531 dexmedetomidine and chloral hydrate sedation for transthoracic echocardiography in infants and
- 532 toddlers: a randomized clinical trial. Pediatr Anesth. 2016;26:266-72.
- 533 27. Li BL, Zhang N, Huang JX, al. e. A comparison of intranasal dexmedetomidine for
- 534 sedation in children administered either by atomiser or by drops. Anaesth. 2016;71:522–8.
- 535 28. Reynolds J, Rogers A, Medellin E, Guzman JA, MF W. A prospective, randomized,
- 536 double-blind trial of intranasal dexmedetomidine and oral chloral hydrate for sedated auditory
- 537 brainstem response (ABR) testing. Pediatr Anesth. 2016;26:286-93.
- 538 29. Li BL, Yuen VM, Song XR, Ye J, Ni J, Huang JX, et al. Intranasal dexmedetomidine
- 539 following failed chloral hydrate sedation in children. Anaesth. 2014;69:240-4.
- 540 30. Yuen VM, Li BL, Cheuk DK, al. e. A randomised controlled trial of oral chloral hydrate
- 541 vs. intranasal dexmedetomidine before computerised tomography in children. Anaesth.
- 542 2017;72:1191–5.
- 543 31. Ghai B, Jain K, Saxena AK, Bhatia N, KS S. Comparison of oral midazolam with
- 544 intranasal dexmedetomidine premedication for children undergoing CT imaging: a randomized,
- 545 double-blind, and controlled study. Pediatr Anesth. 2017;27:37-44.
- 546 32. Tug A, Hanci A, Turk HS, Aybey F, Isil CT, Sayin P, et al. Comparison of two different
- 547 intranasal doses of dexmedetomidine in children for magnetic
- 548 resonance imaging sedation. Pediatr Drugs. 2015;17:479-85.
- 549 33. Zhang W, Wang Z, Song X, Fan Y, Tian H, B L. Comparison of rescue techniques for
- 550 failed chloral hydrate sedation for magnetic resonance imaging scans—additional chloral hydrate
- vs intranasal dexmedetomidine. Pediatr Anesth. 2016;26:273-9.
- Gupta A, Dalvi NP, BA T. Comparison between intranasal dexmedetomidine and
- 553 intranasal midazolam as premedication
- 554 for brain magnetic resonance imaging in pediatric patients: A prospective randomized double
- 555 blind trial. J Anaesthesiol Clin Pharmacol. 2017;33:236-40.
- Gyanesh P, Haldar R, Srivastava D, Agrawal PM, Tiwari AK, Singh PK. Comparison
- 557 between intranasal deximedetomidine and intranasal ketamine as premedication for procedural
- 558 sedation in children undergoing MRI: a double-blind, randomized, placebo-controlled trial.
- 559 Journal of anesthesia. 2014;28(1):12-8.
- 560 36. Ibrahim M. A prospective, randomized, double blinded comparison of intranasal
- 561 dexmedetomodine vs intranasal ketamine in combination with intravenous midazolam for
- 562 procedural sedation in school aged children undergoing MRI. Anesthesia, Essays and
- 563 Researches. 2014;8(2):179-86.
- 564 37. Qiao H, Xie Z, J J. Pediatric premedication: a double-blind randomized trial of
- 565 dexmedetomidine or ketamine alone versus a combination of dexmedetomidine and ketamine.
- 566 BMC Anaesth. 2017;17:158-65.
- 567 38. Xie Z, Shen W, Lin J, Xiao L, Liao M, X G. Sedation effects of intranasal
- 568 dexmedetomidine delivered as sprays versus drops on pediatric response to venous cannulation.
- 569 Am J Emerg Med. 2017;35:1126–30.
- 570 39. Neville DNW, Hayes KR, Ivan Y, McDowell ER, RD P. Double-blind randomized
- 571 controlled trial of intranasal dexmedetomidine versus intranasal

Study: Intranasal dexmedetomidine for laceration repair in children: a dose finding study

Protocol: Dose Finding Study Version 3.5 – November 1, 2019

- 572 midazolam as anxiolysis prior to pediatric laceration repair in the emergency department. Acad
- 573 Emerg Med. 2016;23:910-7.
- Surendar MN, Pandey RK, Saksena AK, Kumar R, Chandra G. A comparative evaluation
- 575 of intranasal dexmedetomidine, midazolam and ketamine for their sedative and analgesic
- 576 properties: a triple blind randomized study. J Clin Pediatr Dent. 2014;38(3):255-61.
- 577 41. Patel V, Singh N, Saksena AK, Singh S, Sonkar SK, SM J. A comparative assessment of
- 578 intranasal and oral dexmedetomidine for procedural sedation in pediatric dental patients. J Indian
- 579 Soc Pedod Prev Dent 2018;36(4):370-5.
- 580 42. Malviya S, Voepel-Lewis T, Burke C, Merkel S, Tait AR. The revised FLACC
- 581 observational pain tool: improved reliability and validity for pain assessment in children with
- 582 cognitive impairment. Pediatric Anesthesia. 2006;16(3):258-65.
- 583 43. Hansen JK, Voss J, Ganatra H, Langner T, Chalise P, Stokes S, et al. Sedation and
- 584 analgesia during pediatric burn dressing change: a survey of American Burn Association centers.
- 585 J Burn Care Res. 2019;40(3):287-93.
- 586 44. Sury M, Bullock I, Rabar S, K D. Sedation for diagnostic and therapeutic procedures in
- 587 children and young people: summary of NICE guidance. BMJ. 2010;341:c6819.
- 588 45. Reynolds J, Rogers A, Capehart S, Manyang P, MF W. Retrospective comparison of
- 589 intranasal dexmedetomidine and oral chloral hydrate for sedated auditory brainstem response
- 590 exams. Hospital Pediatrics. 2016;6(3):166-71.
- 591 46. Cotè CJ, Karl HW, Notterman DA, Wemberg JA, C M. Adverse sedation events in
- 592 pediatrics: analysis of medications used for sedation. Pediatrics. 2000;106:633-44.
- 593 47. Fong CY, Tay CG, Ong LC, NM L. Chloral hydrate as a sedating agent for
- 594 neurodiagnostic procedures in children. Cochrane Database of Systematic Reviews.
- 595 2017;11:CD011786.
- US Food and Drug Safety Administration Safety Communication: FDA review results in
- 597 new warnings about using general anesthetics and sedation drugs in young children and pregnant
- 598 women 2016 [updated March 8, 2018]. Available from: <a href="https://www.fda.gov/drugs/drug-safety-">https://www.fda.gov/drugs/drug-safety-</a>
- 599 and-availability/fda-drug-safety-communication-fda-review-results-new-warnings-about-using-
- 600 general-anesthetics-and.
- 601 49. Koo E, Oshodi T, Meschter C, al e. Neurotoxic effects of dexmedetomidine in fetal
- 602 cynomolgus monkey brains. J Toxicol Sci. 2014;39:251-62.
- Graudins A, Meek R, Egerton-Warburton D, Oakley E, Seith R. The PICHFORK (Pain in
- 604 Children Fentanyl or Ketamine) Trial: A Randomized Controlled Trial Comparing Intranasal
- 605 Ketamine and Fentanyl for the Relief of Moderate to Severe Pain in Children With Limb
- 606 Injuries. Annals of Emergency Medicine. 2015;65(3):248-54. e1.
- 51. Frey TM, Florin TA, Caruso M, Zhang N, Zhang Y, MR M. Effect of intranasal ketamine
- on pain reduction for extremity injuries in children: the PRIME randomized clinical
- 609 trial. JAMA Pediatr. 2019;173(2):140-6.
- 610 52. Anttila M, Penttila J, Helminen A, Vuorilehto L, H S. Bioavailability of
- dexmedetomidine after extravascular doses in healthy subjects. Br J Clin Pharmacol.
- 612 2003;56(6):691-3.
- 613 53. Iirola T, Vilo A, Manner T, Aantaa R, Lahtinen M, Scheinin M, et al. Bioavailability of
- 614 dexmedetomidine after intranasal administration. Eur J Clin Pharmacol. 2011;67:825–31.
- 615 54. Talon MD, Woodson LC, Sherwood ER, Aarsland A, McRae L, T B. Intranasal
- 616 dexmedetomidine premedication is comparable with midazolam in burn children undergoing
- 617 reconstructive surgery. J Burn Care Res. 2009;30(4):599-605.

- Pandey RK, Bahetwar SK, Saksena AK, Chandra G. A comparative evaluation of drops
- 619 versus atomized administration of intranasal ketamine for the procedural sedation of young
- 620 uncooperative pediatric dental patients: A prospective crossover trial. Journal of Clinical
- 621 Pediatric Dentistry. 2011;36(1):79-84.
- 622 56. Ghali AM, Mahfouz AK, M A-B. Preanesthetic medication in children: a comparison of
- 623 intranasal dexmedetomidine versus oral midazolam. Saudi J Anaesth 2011;5:387-91.
- Uusalo P, Jätinvuori H, Löyttyniemi E, Kosola J, T S. Intranasal low-dose
- dexmedetomidine reduces postoperative opioid requirement in patients undergoing hip
- 626 arthroplasty under general anesthesia. J Arthroplasty. 2019.
- 627 58. Aydogan MS, Korkmaz MF, Ozgül U ea. Pain, fentanyl consumption, and delirium in
- 628 adolescents after scoliosis surgery: dexmedetomidine
- 629 vs midazolam. Paediatr Anaesth. 2013;23:446-52.
- 630 59. Prasad SR, Simha PP, AM J. Comparative study between dexmedetomidine and fentanyl
- 631 for sedation during mechanical ventilation in post-operative paediatric cardiac surgical patients.
- 632 Indian J Anaesth. 2012;56:547-52.
- 633 60. Bansal P, Garg S. Effect of adding dexmedetomidine to local anesthetic agents for
- 634 transversus abdominis plane block: a meta-analysis. Clin J Pain. 2019.
- 635 61. Yuen VM, Hui TW, Irwin MG, Yao TJ, Wong GL, MK Y. Optimal timing for the
- 636 administration of intranasal dexmedetomidine for premedication in children. Anaesth.
- 637 2010;65(9):922-9.
- 638 62. Coté CJ, Wilson S, American Academy of Pediatrics, Dentistry AAoP. Guidelines for
- 639 monitoring and management of pediatric patients before, during, and after sedation for diagnostic
- and therapeutic procedures: update 2016, Pediatrics. 2016;138(1):e1-e31.
- 641 63. Yuen VM, Irwin MG, Hui TW, al. e. A double-blind, crossover assessment of the
- 642 sedative and analgesic effects of intranasal dexmedetomidine. Anesth Analg. 2007;105:374-80.
- 643 64. Tobias JD, Berkenbosch JW. Sedation during mechanical ventilation in infants and
- 644 children: dexmedetomidine versus midazolam. South Med J. 2004;97:451-5.
- 645 65. Ewing-Cobbs L, Bloom DR, Prasad MR, Waugh JK, Cox CS Jr, PR S. Assessing
- 646 recovery and disability after physical trauma: the Pediatric Injury Functional Outcome Scale. J
- 647 Pediatr Psychol. 2014;39(6):653-65.
- 648 66. Bhatt M KR, Osmond MH, Krauss B, McAllister JD, Ansermino JM, Evered LM,
- 649 Roback M. Consensus Panel on Sedation Research of Pediatric Emergency Research Canada and
- 650 the Pediatric Emergency Care Applied Research Network. Consensus-based recommendations
- 651 for standardizing terminology and reporting adverse events for emergency department procedural
- 652 sedation and analgesia in children. Ann Emerg Med. 2009;53(4):426-35.e4.
- 653 67. Godwin SA, Burton JH, Gerardo CJ, al. e. Clinical Policy: Procedural Sedation and
- 654 Analgesia in the Emergency Department. Ann Emerg Med. 2014;63(2):247-58.

656 657

655

658

661

- Figure Legends
- 659 Figure 1 legend.
- 660 Reasons for exclusion include adult population and/or intravenous dexmedetomidine
- 662 Figure 2 legend.
- 663 Low risk of bias; Unclear risk of bias; High risk of bias

664 665 Figure 3 legend. 666 CI: Confidence interval; OR: Odds ratio; MD: Mean difference; IN: intranasal 667 668 669 670 671 672 673 674 675 Table 1. Characteristics of included trials 676 Source, trial Age range; Comparisons Measure of Results Summary design, (analysis sample effectiveness of size) sedation country, indication for sedation Cao 2017 3-36 months; IN DXM 2 Proportion with IN DXM 2 Favorable for Parallel mcg/kg 61/71 IN DXM 2 (n=141)"Successful mcg/kg; group RCT (85.9%) versus Oral chloral sedation to mcg/kg versus China hydrate 80 complete the oral chloral oral chloral hydrate 45/70 Ophthalmic mg/kg examination" hydrate 80 (64.3%) mg/kg examination based on the Observer's (p=0.003)Assessment of Alertness/Sedation (OAA/S) score ≤ Chen 2019 6-24 months IN DXM 2 Modified No significant Neutral for IN Parallel Observer's DXM<sub>2</sub> (n=100)mcg/kg; difference in group IN DXM 3 Assessment of mean (SD) mcg/kg versus RCT Alertness/Sedation sedation scores IN DXM 3 mcg/kg China (MOAA/S) score between IN mcg/kg Ophthalmic DXM 2 examination mcg/kg [2.6 (2.1)] and IN DXM 3 mcg/kg [2.7 (1.9)] (p>0.05) IN DXM 2 Gan 2016 5-36 months; Following Proportion with Favorable for IN DXM 2 Parallel failure of "Successful mcg/kg 28/30 (n=60)group RCT oral or rectal ophthalmic (93.3%) versus mcg/kg versus China chloral examination" IN DXM 1 IN DXM 1 based on 4-point mcg/kg 20/30 Ophthalmic hydrate 80 mcg/kg examination Likert scale score (66.7%) mg/kg: of 1 (p=0.02)IN DXM 1 mcg/kg; IN DXM 2

https://mc.manuscriptcentral.com/pediatrics

mcg/kg

| Ghai 2017 Parallel group RCT India IV insertion and CT | 1-6 years;<br>(n=59) | IN DXM 2.5<br>mcg/kg;<br>Oral midazolam<br>0.5<br>mg/kg | Sedation level based on Groningen Distress Rating Scale (IV insertion) and proportion with "adequate sedation" based on Ramsay Sedation Score ≥ 4 (CT) | Intravenous insertion: Significantly lower median (IQR) scores with IN DXM 2.5 mcg/kg [1 (1)] versus oral midazolam 0.5 mg/kg [2 (1)] (p=0.04) Completion of procedure not reported CT: IN DXM 2.5 mcg/kg 20/30 (67%) versus oral midazolam 0.5 mg/kg 7/29 (24%) (p=0.002) | Favorable for<br>IN DXM 2.5<br>mcg/kg versus<br>oral<br>midazolam 0.5<br>mg/kg |
|---|---|---|---|---|---|
| Gupta 2017 Parallel group RCT India IV insertion | 1-8 years;<br>(n=60) | IN DXM 1<br>mcg/kg;<br>IN midazolam<br>0.2<br>mg/kg | Proportion that<br>allowed IV<br>insertion without<br>crying and<br>Observer's<br>Assessment of<br>Alertness/Sedation<br>score ≤ 4 | IN DXM 1<br>mcg/kg 24/30<br>(80%) versus<br>IN midazolam<br>0.2 mg/kg<br>16/30 (53%) | Favorable for<br>IN DXM 1<br>mcg/kg versus<br>IN midazolam<br>0.2 mg/kg |
| Gyanesh 2014 Parallel group RCT India IV insertion | 1-10 years<br>(n=150) | IN DXM 1<br>mcg/kg;<br>IN ketamine 5<br>mg/kg;<br>IN saline | Proportion with satisfactory IV cannulation based on de novo "ease of cannulation score" \( \geq 4 \) | IN DXM 1<br>mcg/kg 20/52<br>(38%) versus<br>IN ketamine 5<br>mg/kg 18/52<br>(35%)<br>(p=0.46)<br>versus IN<br>saline 1/46<br>(2%) (p<0.01<br>for both agents<br>versus saline) | Neutral for IN<br>DXM 1<br>mcg/kg versus<br>IN ketamine 5<br>mg/kg |
| Ibrahim 2014 Parallel group RCT Saudi Arabia IV insertion and MRI | 4-10 years<br>(n=58) | IN DXM 3<br>mcg/kg;<br>IN ketamine 7<br>mg/kg | IV insertion: Proportion with "satisfactory acceptance" based on de novo 4- point scale value > 3 MRI: Sedation failure rate based on the Modified Ramsay Sedation Scale | IV insertion:<br>IN DXM 3<br>mcg/kg 27/29<br>(93%) versus<br>IN ketamine 7<br>mg/kg 27/29<br>(93%)<br>(p=0.45) <sup>1</sup><br>MRI:<br>IN DXM 3<br>mcg/kg 4/29<br>(14%) versus | Neutral for IN<br>DXM 3<br>mcg/kg versus<br>IN ketamine 7<br>mg/kg for both<br>IV insertion<br>and MRI |

| | | | | IN ketamine 7<br>mg/kg 6/29<br>(21%)<br>(p=0.48)<br>All<br>successfully<br>completed<br>MRI | |
|---|---|---|---|---|---|
| Li 2014 Parallel group RCT China Diagnostic procedures <sup>2</sup> | 1 month to 13<br>years<br>(n=213) | Following<br>failure of<br>oral chloral<br>hydrate 50<br>mg/kg:<br>IN DXM 1<br>mcg/kg, 1.5<br>mcg/kg, 2<br>mcg/kg | Adequate sedation<br>based on the<br>Modified<br>Observer's<br>Assessment/<br>Alertness Scale<br>score from 0-3 | IN DXM 1<br>mcg/kg 56/67<br>(84%) versus<br>IN DXM 1.5<br>mcg/kg 66/74<br>(89%) versus<br>IN DXM 2<br>mcg/kg 51/53<br>(96%)<br>(p=0.03³) | Favorable for<br>higher doses of<br>IN DXM |
| Li 2016 Parallel group RCT China Transthoracic echocardio- graphy | 2-36 months<br>(n=280) | IN DXM 3<br>mcg/kg<br>using either a<br>mucosal<br>atomizer device<br>(MAD)<br>or nasal drops | "Successful<br>sedation" based on<br>a University of<br>Michigan<br>Sedation Scale<br>score from 2-4 | IN DXM 3<br>mcg/kg via<br>MAD 113/137<br>(83%) versus<br>drops 120/142<br>(85%)<br>(p=0.57) | Neutral for IN<br>DXM 3<br>mcg/kg via<br>MAD versus<br>drops |
| Miller 2015 Parallel group RCT United States & China Transthoracic echocardio- graphy | 3-36 months<br>(n=150) | IN DXM 2<br>mcg/kg;<br>IN DXM 3<br>mcg/kg;<br>Chloral hydrate<br>70<br>mg/kg | Adequate sedation<br>based on a<br>Ramsay Sedation<br>Score ≥ 3 | IN DXM 2<br>mcg/kg 50/50<br>(100%) versus<br>IN DXM 3<br>mcg/kg (48/50)<br>(96%) versus<br>chloral hydrate<br>70 mg/kg<br>48/50 (96%)<br>(p=0.36) | Neutral for IN<br>DXM 2<br>mcg/kg and 3<br>mcg/kg versus<br>chloral hydrate<br>70 mg/kg |
| Neville 2016 Parallel group RCT United States Laceration repair | 1-5 years (n=38) | IN DXM 2<br>mcg/kg;<br>IN midazolam<br>0.4<br>mg/kg | "Not anxious" at<br>the time of wound<br>washout based on<br>the Yale<br>Preoperative<br>Anxiety Scale<br>score ≤ 30 | IN DXM 2<br>mcg/kg 7/20<br>(35%) versus<br>IN midazolam<br>0.4 mg/kg 1/18<br>(6%) [OR 3;<br>95% CI 1-12]<br>Completion of<br>procedure not<br>reported | Neutral for IN<br>DXM 2<br>mcg/kg versus<br>IN midazolam<br>0.4 mg/kg |

| Patel 2018 Parallel group RCT India Dental procedures | 4-9 years<br>(n=44) | IN DXM 2.5<br>mcg/kg;<br>IN DXM 2<br>mcg/kg;<br>Oral DXM 4<br>mcg/kg;<br>Oral DXM 5<br>mcg/kg | "Safe and successful" based on a de novo 5-point scale for response to treatment and adequate sedation, physiologic parameters, and adverse effects with a value $\leq 2$ | IN DXM 2.5<br>mcg/kg 9/11<br>(82%) versus<br>IN DXM 2<br>mcg/kg 3/11<br>(27%) versus<br>oral DXM 4<br>mcg/kg 0/11<br>(0%) versus<br>oral DXM 5<br>mcg/kg 0/11<br>(0%) (p=0.05³) | Favorable for<br>IN DXM 2.5<br>mcg/kg versus<br>all other<br>comparators |
|---|---|---|---|---|---|
| Qiao 2017<br>Parallel<br>group RCT<br>China<br>Intravenous<br>insertion | 2-5 years<br>(n=135) | IN DXM 2.5<br>mcg/kg;<br>Oral ketamine 6<br>mg/kg;<br>IN DXM 2<br>mcg/kg plus<br>oral ketamine 3<br>mg/kg | "Successful venous cannulation" based on de novo 5-point sedation scale value ≤ 2 | IN DXM 2.5<br>mcg/kg 20/42<br>(47%) versus<br>oral ketamine 6<br>mg/kg 28/41<br>(68%) versus<br>IN DXM 2<br>mcg/kg plus<br>oral ketamine 3<br>mg/kg 33/41<br>(80%)<br>(p=0.006³) | Unfavorable<br>for IN DXM<br>2.5 mg/kg<br>versus<br>combination of<br>IN DXM 2<br>mcg/kg plus<br>oral ketamine 3<br>mg/kg and oral<br>ketamine 6<br>mg/kg |
| Reynolds 2016 Parallel group RCT United States Auditory brainstem response testing | 6 months-8 years<br>(n=85) | IN DXM 3<br>mcg/kg;<br>Chloral hydrate<br>50<br>mg/kg | "Satisfactory sedation" based on ability of audiologist to complete the procedure by placing electrodes within 30 minutes | IN DXM 3<br>mcg/kg 39/44<br>(89%) versus<br>chloral hydrate<br>50 mg/kg<br>27/41 (66%)<br>(p=0.18) | Favorable for<br>IN DXM 3<br>mcg/kg versus<br>chloral hydrate<br>50 mg/kg |
| Surendar 2014 Parallel group RCT India Dental procedures | 4-14 years<br>(n=84) | IN DXM 1.5<br>mcg/kg;<br>IN DXM 1<br>mcg/kg;<br>IN midazolam<br>0.2<br>mg/kg;<br>IN ketamine 5<br>mg/kg | "Satisfactory<br>sedation" for the<br>first 30 minutes of<br>the procedure<br>based on a de<br>novo 5-point scale<br>(4 or 5) | IN DXM 1.5<br>mcg/kg 18/21<br>(86%) versus<br>IN DXM 1<br>mcg/kg 17/21<br>(81%) versus<br>IN midazolam<br>0.2 mg/kg<br>13/21 (62%)<br>versus IN<br>ketamine 5<br>mg/kg 14/21<br>(67%)<br>(p=0.24³) | Neutral for IN<br>DXM 1.5<br>mcg/kg and IN<br>DXM 1<br>mcg/kg versus<br>IN midazolam<br>0.2 mg/kg and<br>IN ketamine 5<br>mg/kg |
| Tug 2015<br>Parallel<br>group RCT<br>Turkey<br>MRI | 1-10 years<br>(n=60) | IN DXM 3<br>mcg/kg;<br>IN DXM 4<br>mcg/kg | "Adequate sedation" based on Ramsay Sedation Score ≥ 5 and no need for rescue sedation for MRI at 45 minutes | IN DXM 3<br>mcg/kg 9/30<br>(30%) versus<br>IN DXM 4<br>mcg/kg 21/30<br>(70%)<br>(p=0.002) | Favorable for<br>IN DXM 4<br>mcg/kg versus<br>IN DXM 3<br>mcg/kg |

| Xie 2015<br>Parallel<br>group RCT<br>China<br>IV insertion | 2-5 years<br>(n=106) | IN DXM 2<br>mcg/kg<br>using mucosal<br>atomizer<br>device;<br>IN DXM 2<br>mcg/kg<br>using drops | Response to IV<br>insertion based on<br>Faces, Legs,<br>Activity, Cry,<br>Consolability<br>(FLACC) score | Median (IQR) FLACC score for IN DXM 2 mcg/kg using mucosal atomizer device was 1 (3.5) versus IN DXM 2 mcg/kg using drops was 3 (4) (p=0.02) All participants had completed IV insertions | Favorable for<br>IN DXM 2<br>mcg/kg using<br>mucosal<br>atomizer<br>device versus<br>IN DXM 2<br>mcg/kg using<br>drops |
|---|---|---|---|---|---|
| Yuen 2017<br>Parallel<br>group RCT<br>China<br>CT | Age range not<br>specified<br>(n=196) | IN DXM 3<br>mcg/kg;<br>Oral chloral<br>hydrate 50mg/kg | "Adequate sedation" based on University of Michigan Sedation Scale score ≥ 3 | IN DXM 3<br>mcg/kg 64/87<br>(74%) versus<br>oral chloral<br>hydrate 81/107<br>(76%)<br>(p=0.74) | Neutral for IN<br>DXM 3<br>mcg/kg versus<br>oral chloral<br>hydrate 50<br>mg/kg |
| Zhang 2016<br>Parallel<br>group RCT<br>China<br>MRI | 1-6 months<br>(n=150) | Following failure of oral chloral hydrate 50 mg/kg: IN DXM 1 mcg/kg; IN DXM 2 mcg/kg; Oral chloral hydrate 25 mg/kg | "Successful sedation" based on the Modified Observer's Assessment of Alertness/Sedation Scale score ≤ 3 | IN DXM 1<br>mcg/kg 47/50<br>(94%) versus<br>IN DXM 2<br>mcg/kg 49/50<br>(98%) versus<br>oral chloral<br>hydrate 25<br>mg/kg 40/50<br>(80%)<br>(p<0.01) | Favorable for<br>IN DXM 1<br>mcg/kg and 2<br>mcg/kg versus<br>oral chloral<br>hydrate 25<br>mg/kg |

CT computed tomography; DXM dexmedetomidine; IN intranasal; IQR interquartile range; IV intravenous; MRI magnetic resonance imaging; RCT randomized controlled trial <sup>1</sup>p value reflects between-group differences in overall 4-point scale Includes computed tomography, auditory brainstem testing; visual evoked potentials <sup>3</sup>p value reflects overall difference between groups

Figure 1. Study Flow Diagram



<u>Figure 2</u>. Review authors' judgements about each risk of bias item presented as percentages across all included studies.



Figure 3. GRADE Evidence Profile

| | | | Certainty: | | | | Manda | stients | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Columb . | SSCSSIICH. | | | Nation 1 | auciis | Effec | <u> </u> | Certainty | Importance |
| Ne of<br>studies | Study design | Risk of bias | Inconsistency | Indirectness | Impression | Other considerations | Intranasal<br>dexmedetomidine | other sedatives | Relative<br>(96% CI) | Absolute<br>(96% CI) | Colony | inpo anc |
| Adequacy o | f Sedation | | | | | | | | | | | |
| 18 | rendomized<br>blais | not serious • | serious » | sefous+ | not serious | none | 1086/1362 (79,7%) | 398/522 (54.0%) | not pooled | see comment | ΦΦ <u></u> ΟΟ | CRITICAL |
| Need for Ad | ditional Sedation | | ' | ' | ' | ' | • | ' | ' | | ' | |
| 5 | rendomized<br>blais | not serious • | not serious | sefous+ | not serious | none | 22/223 (9.9%) | 47/167 (28.1%) | not pooled | see comment | ⊕⊕⊕⊜<br>MODERATE | CRITICAL |
| Onset of Se | dation | | | | | | | | | | | |
| 11 | rendomized<br>blais | sefous 4 | serious * | not serious | not serious | none | IN dexmedetonic | line range 7-31 minutes; | IN comparator range 7- | 44.2 minutes | ФФОО | MPORTANT |
| Duration of | Sedation | | | | | | | | | | | |
| 6 | rendomized<br>blais | sefous 4 | not serious | not serious | not serious | none | IN dexmedetomidin | e range 41-91.5 minutes | ; IN comparator range 7 | 7-85.9 minutes | ⊕⊕⊕○<br>MODERATE | MPORTANT |
| Length of 3 | tay | | | | | | | | | | | |
| 4 | rendomized<br>blais | not serious | not serious | not serious | not serious | none | IN dexmedetonidin | e renge 76.8-156 minute | s; IN comparator range ( | 95-144 minutes | ⊕⊕⊕⊕<br>Нон | IMPORTANT |
| Analgesia | | | | | | • | | | | | | |
| 1 | rendomized<br>triels | not serious | sefous ( | not serious | sefous | none | | ference in the mean (30)<br>g [3.8 (0.8)], IND 1.5 mo<br>and IN ketamine [3.5 | g/kg [3.7 (0.9]], IN mids | | ©Q⊕⊕<br>OQ⊕⊕ | MPORTANT |
| Adverse Eff | tots | | | | | • | • | | | | | |
| 18 | rendomized<br>blais | sefous 44 | not serious | not serious | not serious | none | 67/727 (9.2%) | 98/591 (16.6%) | not pooled | see comment | ⊕⊕⊕○<br>MODERATE | CRITICAL |
| Acceptance | of IN Administrati | on | | | | • | | | | | | |
| 4 | rendomized<br>triels | serious 1 | not serious | not serious | not serious | none | | well accepted by 199/26<br>in due to refusal. One stu-<br>by 42/42 (100%) of | utly reported IN midszola | | ⊕⊕⊕⊜<br>MODERATE | MPORTANT |

CI: Confidence Interval: OR: Odds ratio: MD: Mean difference

#### Explanations

- We chose not to downgreate for allocation concessment (selection bias) because although most brials were judged to have an unclear risk of bias, in all cases this was due to insufficient details provided
   Dignificant heleogeneity (I-squared=70%) partially explained by different comparations

- c. Use of a non-standardized tool to determine level and adequacy of sedation in at least one study limits the degree to which the results can be applied broadly
  d. Use of non-standardized tools to define the onset of sedation was previsient across trials
  e. Downgreded for consistency due to the large range in this outcome, which was in turn likely due to heterogeneity in measurement instruments, dose, and comparators
  f. Unable to assess given only one study reporting this outcome
  g. Total sample size < 200 participants
  h. U et al. was judged to have high risk of bias for incomplete outcome data because 14/67 participants in the IND 2 mogfing arm withdraw post-randomization and did not return to the sedation centre
  l. Burendare et al. did not report adverse effects but reported that signs during sedation that appeared to be within physiologic parameters and the risk of bias was deemed to be unclear
  j. Adverse effects were not defined using standardized or objective criteria
  k. Use of non-standardized tools to assess tolerability of IN sprays limits the degree to which the results can be applied broadly

| Source, trial<br>design,<br>country,<br>indication for<br>sedation | Age<br>range;<br>(analysis<br>sample<br>size) | Comparisons | Measure of<br>effectiveness of<br>sedation | Results | Summary |
|---|---|---|---|---|---|
| Cao 2017<br>Parallel group<br>RCT<br>China<br>Ophthalmic<br>examination | 3-36<br>months;<br>(n=141) | IN DXM 2 mcg/kg;<br>Oral chloral hydrate 80<br>mg/kg | Proportion with "Successful sedation to complete the examination" based on the Observer's Assessment of Alertness/Sedation (OAA/S) score = 4 | IN DXM 2 mcg/kg 61/71 (85.9%)<br>versus oral chiloral hydrate 45/70<br>(64.3%) (p=0.003) | Favorable<br>for IN DXM<br>2 mcg/kg<br>versus oral<br>chloral<br>hydrate 80<br>mg/kg |
| Chen 2019<br>Parallel group<br>RCT<br>China<br>Ophthalmic<br>examination | 6-24<br>months<br>(n=100) | IN DXM 2 mcg/kg;<br>IN DXM 3 mcg/kg | Modified<br>Observer's<br>Assessment of<br>Alertness/Sedation<br>(MOAA/S) score<br>with successful<br>sedation 0-3 | No significant difference in mean (SD) sedation scores between IN DXM 2 mcg/kg [2.6 (2.1)] and IN DXM 3 mcg/kg [2.7 (1.9)] (p=0.05) IND 2 mcg/kg: 49/50 completed all procedures IND 3 mcg/kg: 50/50 completed all procedures | Neutral for<br>IN DXM 2<br>mcg/kg<br>versus IN<br>DXM 3<br>mcg/kg |
| Gan 2016<br>Parallel group<br>RCT<br>China<br>Ophthalmic<br>examination | 5-36<br>months;<br>(n=60) | Following failure of<br>oral or rectal chloral<br>hydrate 80 mg/kg:<br>IN DXM 1 mcg/kg;<br>IN DXM 2 mcg/kg | Proportion with "Successful ophthalmic examination" based on 4-point Likert scale score of 1 | IN DXM 2 mcg/kg 28/30 (93.3%)<br>versus IN DXM 1 mcg/kg 20/30<br>(66.7%) (p=0.02) | Favorable<br>for IN DXM<br>2 mcg/kg<br>versus IN<br>DXM 1<br>mcg/kg |
| Ghai 2017<br>Parallel group<br>RCT<br>India<br>IV insertion<br>and CT | 1-6<br>years;<br>(n=59) | IN DXM 2.5 mcg/kg;<br>Oral midazolam 0.5<br>mg/kg | Sedation level<br>based on<br>Groningen Distress<br>Rating Scale (IV<br>insertion) and<br>proportion with<br>"adequate | Intravenous insertion: Significantly lower median (IQR) scores with IN DXM 2.5 mcg/kg [1 (1)] versus oral midazolam 0.5 mg/kg [2 (1)] (p=0.04) Completion of procedure not reported CT: | Favorable<br>for IN DXM<br>2.5 mcg/kg<br>versus oral<br>midazolam<br>0.5 mg/kg |

| | | | sedation" based on<br>Ramsay Sedation<br>Score ≥ 4 (CT) | IN DXM 2.5 mcg/kg 20/30 (67%)<br>versus oral midazolam 0.5 mg/kg 7/29<br>(24%) (p=0.002) | |
|---|---|---|---|---|---|
| Gupta 2017<br>Parallel group<br>RCT<br>India<br>IV insertion | 1-8<br>years;<br>(n=60) | IN DXM 1 mcg/kg;<br>IN midazolam 0.2<br>mg/kg | Proportion that<br>allowed IV<br>insertion without<br>crying and<br>Observer's<br>Assessment of<br>Alertness/Sedation<br>score ≤ 4 | IN DXM 1 mcgkg 24/30 (80%) versus<br>IN midszolam 0.2 mg/kg 16/30 (53%) | Favorable<br>for IN DXM<br>1 mcg/kg<br>versus IN<br>midazolam<br>0.2 mg/kg |
| Gyanesh<br>2014<br>Parallel group<br>RCT<br>India<br>IV insertion | 1-10<br>years<br>(n=150) | IN DXM 1 mcg/kg;<br>IN ketumine 5 mg/kg;<br>IN saline | Proportion with satisfactory IV cannulation based on the novo "ease of cannulation score" 4 | IN DXM 1 mcg/kg 20/52 (38%) versus<br>IN ketamine 5 mg/kg 18/52 (35%)<br>(p=0.46) versus IN saline 1/46 (2%)<br>(p=0.01 for both agents versus saline) | Neutral for<br>IN DXM 1<br>mcg/kg<br>versus IN<br>ketamine 5<br>mg/kg |
| Ibrahim 2014<br>Parallel group<br>RCT<br>Saudi Arabia<br>IV insertion<br>and MRI | 4-10<br>years<br>(n=58) | IN DXM 3 mcg/kg;<br>IN ketamine 7 mg/kg | IV insertion: Proportion with "satisfactory acceptance" based on de novo 4-point scale value ≥ 3 MRI: Sedation failure rate based on the Modified Ramsay Sedation Scale | IV insertion: IN DXM 3 mcg/kg 27/29 (93%) versus IN ketamine 7 mg/kg 27/29 (93%) (p=0.45)) MRI: IN DXM 3 mcg/kg 4/29 (14%) versus IN ketamine 7 mg/kg 6/29 (21%) (p=0.48) All successfully completed MRI | Neutral for<br>IN DXM 3<br>mcg/kg<br>versus IN<br>ketamine 7<br>mg/kg for<br>both IV<br>insertion and<br>MRI |

| Li 2014<br>Parallel group<br>RCT<br>China<br>Diagnostic<br>procedures <sup>2</sup> | 1 month<br>to 13<br>years<br>(n=213) | Following failure of<br>oral chloral hydrate 50<br>mg/kg:<br>DV DXM 1 mcg/kg, 1.5<br>mcg/kg, 2 mcg/kg | Adequate sedation<br>based on the<br>Modified<br>Observer's<br>Assessment/<br>Alertness Scale<br>score from 0-3 | IN DXM 1 mcg/kg 56/67 (84%) versus<br>IN DXM 1.5 mcg/kg 66/74 (89%)<br>versus IN DXM 2 mcg/kg 51/53 (96%)<br>(p=0.03 <sup>3</sup> ) | Favorable<br>for higher<br>doses of IN<br>DXM |
|---|---|---|---|---|---|
| Li 2016<br>Parallel group<br>RCT<br>China<br>Transthoracic<br>echocardio-<br>graphy | 2-36<br>months<br>(n=280) | IN DXM 3 mcg/kg<br>using either a mucosal<br>atomizer device (MAD)<br>or nasal drops | "Successful<br>sedation" based on<br>a University of<br>Michigan Sedation<br>Scale score from 2-<br>4 | IN DXM 3 mcg/kg via MAD 113/137<br>(83%) versus drops 120/142 (85%)<br>(p=0.57) | Neutral for<br>IN DXM 3<br>mcg/kg via<br>MAD versus<br>drops |
| Miller 2015 Parallel group RCT United States & China Transtheracic echocardio- graphy | 3-36<br>months<br>(n=150) | IN DXM 2 mcg/kg;<br>IN DXM 3 mcg/kg;<br>Chloral hydrate 70<br>mg/kg | Adequate sedation<br>based on a Ramsay<br>Sedation Score ≥ 3 | IN DXM 2 mcg/kg 50/50 (100%) versus<br>IN DXM 3 mcg/kg (48/50) (96%) versus<br>chloral hydrate 70 mg/kg 48/50 (96%)<br>(p=0.36) | Neutral for<br>IN DXM 2<br>mcg/kg and<br>3 mcg/kg<br>versus<br>chloral<br>hydrate 70<br>mg/kg |
| Neville 2016<br>Parallel group<br>RCT<br>United States<br>Laceration<br>repair | 1-5 years<br>(n=38) | IN DXM 2 mcg/kg;<br>IN midazolam 0.4<br>mg/kg | "Not anxious" at<br>the time of wound<br>washout based on<br>the Yale<br>Preoperative<br>Anxiety Scale<br>score = 30 | IN DXM 2 mcg/kg 7/20 (35%) versus<br>IN midszolam 0.4 mg/kg 1/18 (6%) [OR<br>3; 95% CI 1-12]<br>Completion of procedure not reported | Neutral for<br>IN DXM 2<br>mcg/kg<br>verus IN<br>midazolam<br>0.4 mg/kg |

| Parel 2018<br>Parellel group<br>RCT<br>India<br>Dental<br>procedures | 4-9 years<br>(a=44) | IN DXM 2.5 mcg/kg;<br>IN DXM 2 mcg/kg;<br>Oral DXM 4 mcg/kg;<br>Oral DXM 5 mcg/kg | "Safe and successful" based on a de novo 5-point scale for response to treatment and adequate sedation, physiologic parameters, and adverse effects with a value \( \sigma 2\) | IN DXM 2.5 mcg/kg 9/11 (82%) versus<br>IN DXM 2 mcg/kg 3/11 (27%) versus<br>oral DXM 4 mcg/kg 0/11 (0%) versus<br>oral DXM 5 mcg/kg 0/11 (0%) (p=0.05°) | Favorable<br>for IN DXM<br>2.5 mcg/kg<br>versus all<br>other<br>comparators |
|---|---|---|---|---|---|
| Qiao 2017<br>Parallel group<br>RCT<br>China<br>Intravenous<br>insertion | 2-5 years<br>(n=135) | DV DXM 2.5 mcg/kg;<br>Oral ketamine 6 mg/kg;<br>DV DXM 2 mcg/kg plus<br>oral ketamine 3 mg/kg | "Successful venous cammilation" based on de novo 5-point sedation scale value ≤ 2 | IN DXM 2.5 mcg/kg 20/42 (47%)<br>versus oral ketamine 6 mg/kg 28/41<br>(68%) versus IN DXM 2 mcg/kg plus<br>oral ketamine 3 mg/kg 33/41 (80%)<br>(p=0.006%) | Unfavorable<br>for IN DXM<br>2.5 mg/kg<br>vervus<br>combination<br>of IN DXM<br>2 mcg/kg<br>plus oral<br>ketamine 3<br>mg/kg and<br>oral<br>ketamine 6<br>mg/kg |
| Reynolds<br>2016<br>Parallel group<br>RCT<br>United States<br>Auditory<br>brainstem<br>response<br>testing | 6<br>months-8<br>years<br>(n=85) | IN DXM 3 mcg/kg;<br>Chloral hydrate 50<br>mg/kg | "Satisfactory sedation" based on ability of audiologist to complete the procedure by placing electrodes within 30 minutes | IN DXM 3 mcg/kg 39/44 (89%) versus<br>chloral hydrate 50 mg/kg 27/41 (66%)<br>(p=0.18) | Favorable<br>for IN DXM<br>3 mcg/kg<br>versus<br>chloral<br>hydrate 50<br>mg/kg |

| Surendar<br>2014<br>Parallel group<br>RCT<br>India<br>Dental<br>procedures | 4-14<br>years<br>(n=84) | IN DXM 1.5 mcg/kg;<br>IN DXM 1 mcg/kg;<br>IN midazolam 0.2<br>mg/kg;<br>IN ketamine 5 mg/kg | "Satisfactory sedation" for the first 30 minutes of the procedure based on a de novo 3-point scale (4 or 5) | IN DXM 1.5 mcg/kg 18/21 (86%) versus IN DXM 1 mcg/kg 17/21 (81%) versus IN midazolam 0.2 mg/kg 13/21 (62%) versus IN ketamine 5 mg/kg 14/21 (67%) (p=0.24*) | Neutral for<br>IN DXM 1.5<br>mcg/kg and<br>IN DXM 1<br>mcg/kg<br>versus IN<br>midazolam<br>0.2 mg/kg<br>and IN<br>ketamine 5<br>mg/kg |
|---|---|---|---|---|---|
| Tug 2015<br>Parallel group<br>RCT<br>Turkey<br>MRI | 1-10<br>years<br>(n=60) | IN DXM 3 mcg/kg;<br>IN DXM 4 mcg/kg | "Adequate sedation" based on Ramsay Sedation Score ≥ 5 and no need for rescue sedation for MRI at 45 minutes | IN DXM 3 mcg/kg 9/30 (30%) versus<br>IN DXM 4 mcg/kg 21/30 (70%)<br>(p=0.002) | Favorable<br>for IN DXM<br>4 mcg/kg<br>verus IN<br>DXM 3<br>mcg/kg |
| Xie 2015<br>Parallel group<br>RCT<br>China<br>IV insertion | 2-5 years<br>(n=106) | IN DXM 2 mcg/kg<br>using muco-sal stomizer<br>device;<br>IN DXM 2 mcg/kg<br>using drops | Response to IV<br>insertion based on<br>Faces, Legs,<br>Activity, Cry,<br>Consolability<br>(FLACC) score | Median (IQR) FLACC score for IN<br>DXM 2 mcg/kg using nuccotal atomizer<br>device was 1 (3.5) yearus IN DXM 2<br>mcg/kg using drops was 3 (4) (p=0.02)<br>All participants had completed IV<br>insertions | Favorable<br>for IN DXM<br>2 mcg/kg<br>using<br>mucosal<br>atomizer<br>device<br>versus IN<br>DXM 2<br>mcg/kg<br>using drops |
| Yuen 2017<br>Parallel group<br>RCT<br>China<br>CT | Age<br>range not<br>specified<br>(n=196) | IN DXM 3 mcg/kg;<br>Oral chloral hydrate 50<br>mg/kg | "Adequate sedation" based on University of Michigan Sedation Scale score ≥ 3 | IN DXM 3 mcg/kg 64/87 (74%) versus<br>oral chloral hydrate 81/107 (76%)<br>(p=0.74) | Neutral for<br>IN DXM 3<br>mcg/kg<br>versus oral<br>chloral<br>hydrate 50<br>mg/kg |

| Zhang 20 | 16 1-6 | Following failure of | "Successful | IN DXM 1 mcg/kg 47/50 (94%) versus | Favorable |
|---|---|---|---|---|---|
| Parallel g | roup months | oral chloral hydrate 50 | sedation" based on | IN DXM 2 mcg/kg 49/50 (98%) versus | for IN DXM |
| RCT | (n=150) | mg/kg: | the Modified | oral chloral hydrate 25 mg/kg 40/50 | 1 mcg/kg |
| China | | | Observer's | (80%) (p=0.01) | and 2 |
| MRI | | IN DXM 1 mcg/kg; | Assessment of | | mcg/kg |
| 1 | | IN DXM 2 mcg/kg; | Alertness/Sedation | | versus oral |
| 1 | | Oral chloral hydrate 25 | Scale score <u>&lt;</u> 3 | | chloral |
| 1 | | mg/kg | | | hydrate 25 |
| | | | | | mg/kg |

CT computed tomography; DXM dexised etomidine; IN intranasal; IQR interquartile range; IV intravenous; MRI magnetic resonance imaging; RCT randomized controlled trial

<sup>&</sup>lt;sup>1</sup>P value reflects between-group differences in overall 4-point scale

Includes computed tomography, auditory brainstem testing; visual evoked potentials

<sup>&</sup>lt;sup>3</sup>P value reflects overall difference between groups



### PRISMA 2009 Checklist

| Section/topic | # | Checklist item | Reported on page # |
|---|---|---|---|
| TITLE | | | |
| Title | 1 | Identify the report as a systematic review, meta-analysis, or both. | Title<br>page |
| ABSTRACT | | | |
| Structured summary | 2 | Provide a structured summary including, as applicable: background; objectives; data sources; study eligibility criteria, participants, and interventions; study appraisal and synthesis methods; results; limitations; conclusions and implications of key findings; systematic review registration number. | 2-3 |
| INTRODUCTION | | | |
| Rationale | 3 | Describe the rationale for the review in the context of what is already known. | 4 |
| Objectives | 4 | Provide an explicit statement of questions being addressed with reference to participants, interventions, comparisons, outcomes, and study design (PICOS). | 4 |
| METHODS | | | |
| Protocol and registration | 5 | Indicate if a review protocol exists, if and where it can be accessed (e.g., Web address), and, if available, provide registration information including registration number. | 5 |
| Eligibility criteria | 6 | Specify study characteristics (e.g., PICOS, length of follow-up) and report characteristics (e.g., years considered, language, publication status) used as criteria for eligibility, giving rationale. | 5 |
| Information sources | 7 | Describe all information sources (e.g., databases with dates of coverage, contact with study authors to identify additional studies) in the search and date last searched. | 5-6 |
| Search | 8 | Present full electronic search strategy for at least one database, including any limits used, such that it could be repeated. | Appendix |
| Study selection | 9 | State the process for selecting studies (i.e., screening, eligibility, included in systematic review, and, if applicable, included in the meta-analysis). | 6 |
| Data collection process | 10 | Describe method of data extraction from reports (e.g., piloted forms, independently, in duplicate) and any processes for obtaining and confirming data from investigators. | 6 |
| Data items | 11 | List and define all variables for which data were sought (e.g., PICOS, funding sources) and any assumptions and simplifications made. | 6 |
| Risk of bias in individual studies | 12 | Describe methods used for assessing risk of bias of individual studies (including specification of whether this was done at the study or outcome level), and how this information is to be used in any data synthesis. | 6 |
| Summary measures | 13 | State the principal summary measures (e.g., risk ratio, difference in means). | 7 |

https://mc.manuscriptcentral.com/pediatrics

57

### INTERNAL PROPERTY.

### PRISMA 2009 Checklist

| 14 | Describe the methods of handling data and combining results of studies, if done, including measures of consistency (e.g., $I^2$ ) for each meta-analysis. | 7 |
|---|---|---|
| | Page 1 of 2 | • |
| # | Checklist item | Reported on page # |
| 15 | Specify any assessment of risk of bias that may affect the cumulative evidence (e.g., publication bias, selective reporting within studies). | 7 |
| 16 | Describe methods of additional analyses (e.g., sensitivity or subgroup analyses, meta-regression), if done, indicating which were pre-specified. | 7 |
| 17 | Give numbers of studies screened, assessed for eligibility, and included in the review, with reasons for exclusions at each stage, ideally with a flow diagram. | 8 |
| 18 | For each study, present characteristics for which data were extracted (e.g., study size, PICOS, follow-up period) and provide the citations. | Table 1 |
| 19 | Present data on risk of bias of each study and, if available, any outcome level assessment (see item 12). | Figure 2 |
| 20 | For all outcomes considered (benefits or harms), present, for each study: (a) simple summary data for each intervention group (b) effect estimates and confidence intervals, ideally with a forest plot. | Table 1 |
| 21 | Present results of each meta-analysis done, including confidence intervals and measures of consistency. | Figure 4 |
| 22 | Present results of any assessment of risk of bias across studies (see Item 15). | Figure 3 |
| 23 | Give results of additional analyses, if done (e.g., sensitivity or subgroup analyses, meta-regression [see Item 18]). | 9-10 |
| 24 | Summarize the main findings including the strength of evidence for each main outcome; consider their relevance to key groups (e.g., healthcare providers, users, and policy makers). | 13-16 |
| 25 | Discuss limitations at study and outcome level (e.g., risk of bias), and at review-level (e.g., incomplete retrieval of identified research, reporting bias). | 16 |
| 26 | Provide a general interpretation of the results in the context of other evidence, and implications for future research. | 16 |
| FUNDING | | |
| 27 | Describe sources of funding for the systematic review and other support (e.g., supply of data); role of funders for the systematic review. | n/a |
| | # 15 16 17 18 19 20 21 22 23 24 25 26 | (e.g., I²) for each meta-analysis. Page 1 of 2 # Checklist item 15 Specify any assessment of risk of bias that may affect the cumulative evidence (e.g., publication bias, selective reporting within studies). 16 Describe methods of additional analyses (e.g., sensitivity or subgroup analyses, meta-regression), if done, indicating which were pre-specified. 17 Give numbers of studies screened, assessed for eligibility, and included in the review, with reasons for exclusions at each stage, ideally with a flow diagram. 18 For each study, present characteristics for which data were extracted (e.g., study size, PICOS, follow-up period) and provide the citations. 19 Present data on risk of bias of each study and, if available, any outcome level assessment (see item 12). 20 For all outcomes considered (benefits or harms), present, for each study: (a) simple summary data for each intervention group (b) effect estimates and confidence intervals, ideally with a forest plot. 21 Present results of each meta-analysis done, including confidence intervals and measures of consistency. 22 Present results of any assessment of risk of bias across studies (see Item 15). 23 Give results of additional analyses, if done (e.g., sensitivity or subgroup analyses, meta-regression [see Item 16]). 24 Summarize the main findings including the strength of evidence for each main outcome; consider their relevance to key groups (e.g., healthcare providers, users, and policy makers). 25 Discuss limitations at study and outcome level (e.g., risk of bias), and at review-level (e.g., incomplete retrieval of identified research, reporting bias). 26 Provide a general interpretation of the results in the context of other evidence, and implications for future research. |

44 From: Moher D, Liberati A, Tetziaff J, Altman DG, The PRISMA Group (2009). Preferred Reporting Items for Systematic Reviews and Meta-Analyses: The PRISMA Statement. PLoS Med 6(6): e1000097. https://mc.manuscriptcentral.com/pediatrics

Search as of July 26, 2019

| # | Query | Results |
|---|---|---|
| S38 | \$36 AND \$37 | 39 |
| \$37 | S13 OR S14 OR S15 OR S16 OR S17 OR S18 OR S19 OR S20 OR S21 OR S22 OR S23 OR S24 OR S25 OR S26 OR S27 OR S28 OR S29 OR S30 OR S31 OR S32 OR S33 OR S34 OR S35 | 2,817 |
| \$36 | S1 OR S2 OR S3 OR S4 OR S5 OR S6 OR S7 OR S8 OR S9 OR S10 OR S11 OR S12 | 1,566 |
| \$35 | (MH "Administration, Intranasal") | 2,371 |
| S34 | medication*, nasal | 80 |
| S33 | nasal medication* | 80 |
| \$32 | medication*, intra-nasal | 0 |
| S31 | intra-nasal medication* | 0 |
| S30 | medication*, intranasal | 49 |
| S29 | intranasal medication* | 49 |
| S28 | instillation*, nasal | 22 |
| S27 | nasal instillation* | 22 |
| S26 | instillation*, intra-nasal | 0 |
| S25 | intra-nasal instillation* | 0 |
| S24 | instillation*, intranasal | 27 |
| S23 | intranasal instillation | 27 |
| S22 | administration*, nasal | 301 |
| S21 | nasal administration* | 301 |
| S20 | intra-nasal drug administration* | 0 |
| S19 | intra-nasal administration* | 2 |
| S18 | drug administration*, intra-nasal | 0 |
| S17 | administration*, intra-nasal | 0 |
| S16 | intranasal drug administration* | 23 |
| S15 | intranasal administration* | 2,517 |
| S14 | drug administration*, intranasal | 27 |
| S13 | administration*, intranasal | 2,517 |

| S12 | sileo | 1 |
|-----|--------------------------------|-------|
| S11 | sedadex | 0 |
| S10 | primadex | 0 |
| S9 | dexdor | 3 |
| \$8 | dexdomitor | 0 |
| S7 | cepedex | 0 |
| S6 | precedex | 14 |
| \$5 | "mpv1440" | 0 |
| S4 | hydrochloride, dexmedetomidine | 13 |
| S3 | "mpv 1440" | 0 |
| S2 | dexmedetomidine hydrochloride | 13 |
| S1 | "Dexmedetomidine" | 1,564 |

### Database(s): Embase Classic+Embase 1947 to 2019 July 25

Search Strategy: # Searches Results 9901 1 dexmedetomidine/ 2 dexmedetomidine.mp. 10149 3 dexmedetomidine hydrochloride.mp. 95 4 hydrochloride, dexmedetomidine.mp. 3 5 mpv 1440.mp. 4 0 6 mpv1440.mp. 7 precedes.mp. 450 8 cepedex.mp. 0 9 dexdomitor.mp. 123 10 dexdor.mp. 41 2 11 primades.mp. 12 sedadex.mp. 0 6 13 sileo.mp. 14 intranasal drug administration/ 14768 84 15 administration\*, intranasal.mp. 16 drug administration\*, intranasal.mp.

| 17 | intranasal administration*.mp. | 4312 |
|---|---|---|
| 18 | intranasal drug administration*.mp. | 39833 |
| 19 | administration*, intra-nasal.mp. | 3 |
| 20 | drug administration*, intra-nasal.mp. | 1 |
| 21 | intra-nasal administration*.mp. | 47 |
| 22 | intra-nasal drug administration*.mp. | 0 |
| 23 | nasal administration*.mp. | 1394 |
| 24 | administration*, nasal.mp. | 29 |
| 25 | intranasal instillation*.mp. | 977 |
| 26 | instillation*, intranasal.mp. | 3 |
| 27 | intra-nasal instillation*.mp. | 18 |
| 28 | instillation*, intra-nasal.mp. | 0 |
| 29 | nasal instillation*.mp. | 361 |
| 30 | instillation*, nasal.mp. | 3 |
| 31 | intranasal medication*.mp. | 94 |
| 32 | medication*, intranasal mp. | 11 |
| 33 | intra-nasal medication*.mp. | 1 |
| 34 | medication*, intra-nasal mp. | 0 |
| 35 | nasal medication* mp. | 73 |
| 36 | medication*, nasal.mp. | 21 |
| 37 | 1 or 2 or 3 or 4 or 5 or 6 or 7 or 8 or 9 or 10 or 11 or 12 or 13 | 10153 |
| 38 | 14 or 15 or 16 or 17 or 18 or 19 or 20 or 21 or 22 or 23 or 24 or 25 or 26 or 27 or 28 or 29 or 30 or 31 or 32 or 33 or 34 or 35 or 36 | 42030 |
| 39 | 37 and 38 | 269 |

### Database(s): Ovid MEDLINE(R) ALL 1946 to July 25, 2019 Search Strategy:

| Jem | uch Stategy. | |
|-----|------------------------------------|---------|
| # | Searches | Results |
| 1 | dexmedetomidine/ | 3137 |
| 2 | dexmedetomidine mp. | 5317 |
| 3 | dexmedetomidine hydrochloride mp. | 60 |
| 4 | hydrochloride, dexmedetomidine.mp. | 1 |

| 5 | mpv 1440.mp. | 3 |
|----|---------------------------------------|-------|
| 6 | mpv1440.mp. | 0 |
| 7 | precedex.mp. | 31 |
| 8 | cepedex.mp. | 0 |
| 9 | desdomitor.mp. | 1 |
| 10 | dexdor.mp. | 8 |
| 11 | primadev.mp. | 0 |
| 12 | sedadex.mp. | 0 |
| 13 | sileo.mp. | 2 |
| 14 | administration*, intranasal mp. | 14057 |
| 15 | drug administration*, intranasal mp. | 1 |
| 16 | intranasal administration*mp. | 3262 |
| 17 | intranasal drug administration*.mp. | 45 |
| 18 | administration*, intra-nasal mp. | 0 |
| 19 | drug administration*, intra-nasal mp. | 0 |
| 20 | intra-nasal administration*.mp. | 28 |
| 21 | intra-nasal drug administration*.mp. | 0 |
| 22 | nasal administration* mp. | 985 |
| 23 | administration*, nasal.mp. | 24 |
| 24 | intranasal instillation* mp. | 676 |
| 25 | instillation*, intranasal.mp. | 2 |
| 26 | intra-nasal instillation*.mp. | 10 |
| 27 | instillation*, intra-nasal.mp. | 0 |
| 28 | nasal instillation*.mp. | 234 |
| 29 | instillation*, nasal.mp. | 3 |
| 30 | intranasal medication*.mp. | 67 |
| 31 | medication*, intranasal mp. | 7 |
| 32 | intra-nasal medication* mp. | 1 |
| 33 | medication*, intra-nasal mp. | 0 |
| 34 | nasal medication* mp. | 55 |
| 35 | medication*, nasal.mp. | 13 |
| _ | | _ |

| 36 | Administration, Intranasal/ | 14038 |
|---|---|---|
| 37 | 1 or 2 or 3 or 4 or 5 or 6 or 7 or 8 or 9 or 10 or 11 or 12 or 13 | 5323 |
| 38 | 14 or 15 or 16 or 17 or 18 or 19 or 20 or 21 or 22 or 23 or 24 or 25 or 26 or 27 or 28 or 29 or 30 or 31 or 32 or 33 or 34 or 35 or 36 | 16415 |
| 39 | 37 and 38 | 96 |

Scopus: 301 results

ALL((Dexmedetomidine OR "dexmedetomidine hydrochloride" OR "hydrochloride, dexmedetomidine" OR "mpv 1440" OR mpv-1440 OR mpv1440 OR precedex OR cepedex OR dexdomitor OR dexdor OR primadex OR sedadex OR sileo) AND ("administration, intranasal" OR "administrations, intranasal" OR "drug administration, intranasal" OR "drug administrations, intranasal" OR "intranasal administration" OR "intranasal administrations" OR "intranasal drug administration" OR "intranasal drug administrations" OR "administration, intra-nasal" OR "administrations, intra-nasal" OR "drug administration, intra-nasal" OR "drug administrations, intra-nasal" OR "intra-nasal administration" OR "intra-nasal administrations" OR "intra-nasal drug administration" OR "intra-nasal drug administrations" OR "nasal administration" OR "nasal administrations" OR "administration, nasal" OR "administrations, nasal" OR "intranasal instillation" OR "intranasal instillations" OR "instillation, intranasal" OR "instillations, intranasal" OR "intra-nasal instillation" OR "intra-nasal instillations" OR "instillation, intranasal" OR "instillations, intra-nasal" OR "nasal instillation" OR "nasal instillations" OR "instillation, nasal" OR "instillations, nasal" OR "intranasal medication" OR "intranasal medications" OR "medication, intranasal" OR "medications, intranasal" OR "intra-nasal medication" OR "intra-nasal medications" OR "medication, intra-nasal" OR "medications, intranasal" OR "nasal medication" OR "nasal medications" OR "medication, nasal" OR "medications, nasal"))

#### Web of Science: 31 results

TS=((Dexmedetomidine OR "dexmedetomidine hydrochloride" OR "hydrochloride, dexmedetomidine" OR "mpv 1440" OR mpv-1440 OR mpv1440 OR precedex OR cepedex OR dexdomitor OR dexdor OR primadex OR sedadex OR sileo) AND ("administration, intranasal" OR "administration, intranasal" OR "drug administration, intranasal" OR "drug administrations, intranasal or "intranasal drug administration" OR "intranasal drug administration" OR "administration, intra-nasal" OR "drug administration, intra-nasal" OR "drug administration, intra-nasal" OR "drug administration, intra-nasal" OR "intra-nasal drug administration" OR "intra-nasal administration" OR "intra-nasal drug administration" OR "intra-nasal drug administration" OR "nasal administration" OR "nasal administration" OR "intra-nasal instillation" OR "intra-nasal instillation, intranasal" OR "instillation, intranasal" OR "intra-nasal instillation, intranasal" OR "instillation, intranasal" OR "intranasal" OR "int

nasal" OR "instillations, intra-nasal" OR "nasal instillation" OR "nasal instillations" OR "instillation, nasal" OR "instillations, nasal" OR "intranasal medication" OR "intranasal medications" OR "medication, intranasal" OR "medications, intra-nasal" OR "intra-nasal medications" OR "intra-nasal medications" OR "medication, intra-nasal" OR "medications, intra-nasal" OR "nasal medication" OR "nasal medications" OR "medication, nasal" OR "medications, nasal"))

Timespan: All years. Indexes: SCI-EXPANDED, SSCI, A&HCI, CPCI-S, CPCI-SSH, ESCI.

#### GRAY LITERATURE SEARCH

Clinical Trials Registries

Search: Dexmedetomidine AND (intranasal OR intra-nasal)

UK Clinical Trials Gateway

0 Results

ISRCTN Register

0 Results

HSRProj

0 Results

NIH Reporter

0 Results

PhRMA Clinical Study Results Database

0 Results

Eli Lilly and Company Clinical Trial Registry

0 Results

Roche Clinical Study Register

0 Results

GlaxoSmithKline Clinical Study Register

0 Results

ClinicalTrials.gov

8 Results

Study 1:

The Clinical Research of Intranasal Dexmedetomidine Used in Plastic Title:

Surgery of Children

Recruitment: Unknown status No Results Available Study Results:

The Efficacy and Safety of Intranasal Dexmedetomidine

Conditions: Interventions: Drug: Normal saline,1 milliliter|Drug: Dexmedetomidine 1 µg.kg-1,1 milliliter Drug: Dexmedetomidine 2µg.kg-1,1 milliliter Drug: Anesthesia induction, 8%

sevoflurane|Drug: Anesthesia maintenance, 2%~3% sevoflurane,fentanyl https://ClinicalTrials.gov/show/NCT02222636 URL:

Study 2:

Title: Efficacy and Optimal Dose Selection of Intranasal Dexmedetomidine During

Breast Lumpectomy Under Local Anaesthesia

Recruitment: Completed
Study Results: No Results Available

Study Results: No Results Available
Conditions: Intranasal Dexmedetomidine Breast Cancer Local Anaesthesia
Drug: 0.9% saline|Drug: dexmedetomidine 1µg.kg-1|Drug:

dexmedetomidine 1.5µg.kg-1|Drug: Dexmedetomidine 2µg.kg-1 URL: https://ClinicalTrials.gov/show/NCT02675049

Study 3:

Title: Safety and Efficacy of Intranasal Dexmedetomidine

Recruitment: Not yet recruiting

Study Results: No Results Available
Conditions: Safety and Efficacy of Intranasal Dexmedetomidine

Interventions: Drug: Dexmedetomidine Drug: Midazolam Hydrochloride Drug: Nitrous

Oxide

URL: https://ClinicalTrials.gov/show/NCT02985697

Study 4:

Title: Intranasal Dexmedetomidine Sedation in Children for Non-painful

Procedures

Not yet recruiting Recruitment: Study Results: No Results Available Conditions: Dexmedetomidine|Sedation Interventions: Drug: Intranasal dexmedetomidine

URL: https://ClinicalTrials.gov/show/NCT03220880

Study 5:

Title: Sedation and Physiological Effects of Intranasal Dexmedetomidine in Severe

COPD

Recruitment: Completed

Study Results: No Results Available

Conditions: COPD|Sedation|Dexmedetomidine

Interventions: Drug: Intranasal dexemdetomidine (IN-DEX) URL: https://ClinicalTrials.gov/show/NCT02211118

Study 6:

Recruitment: Completed
Study Results: Has Results
Conditions: Benign Neoplasm of Vocal Fold - Glottis
URL: Dexmedetomidine Premedication
Completed
Has Results
Benign Neoplasm of Vocal Fold - Glottis
Drug: Dexmedetomidine URL: https://ClinicalTrials.gov/show/NCT02108171

Study 7:

Intranasal Dexmedetomidine Sedation for Pediatric CT Imaging Title:

Recruitment: Unknown status

Study Results: No Results Available
Conditions: Traumatic Brain Injury|Children
Interventions: Drug: Dexmedetomidine

URL: https://ClinicalTrials.gov/show/NCT01900405

Study 8:

Title: Bioavailability of Dexmedetomidine After Intranasal Administration

Recruitment: Completed

No Results Available Study Results:

Conditions: Sedation

Interventions: Drug: Intravenous dexmedetomidine Drug: Intranasal dexmedetomidine

URL: https://ClinicalTrials.gov/show/NCT00837187

Study 9:

Title: Intranasal Dexmedetomidine vs Intranasal Midazolam as Anxiolysis Prior to

Pediatric Laceration Repair

Recruitment: Completed Study Results: Has Results Conditions: Laceration|Anxiety

Interventions: Drug: Dexmedetomidine|Drug: Midazolam URL: https://ClinicalTrials.gov/show/NCT02168439

Study 10:

Intranasal Dexmedetomidine vs Midazolam-ketamine Combination for

Premedication of Pediatric Patients Recruitment: Completed

Study Results: No Results Available

Conditions: Premedication|Oculocardiac Reflex
Interventions: Drug: Dexmedetomidine|Drug: Ketamine
URL: https://ClinicalTrials.gov/show/NCT02072083

Study 11:

Title: Intranasal Dexmedetomidine Sedation During Intra-articular Joint Injections

in Pediatric Population

Recruitment: Recruiting

Study Results: No Results Available
Conditions: Juvenile Idiopathic Arthritis|Joint Inflammation
Interventions: Drug: Dexmedetomidine|Drug: Sedatives/Hypnotics,Other
URL: https://ClinicalTrials.gov/show/NCT03069638

Study 12: Placebo Controlled Evaluation of Sedation and Physiological Response to Title:

Intranasal Dexmedetomidine in Severe COPD Recruitment: Not yet recruiting
Study Results: No Results Available
Conditions: COPD
Interventions: Drug: IN-DEX 1.0 mcg/kg, intranasal saline|Drug: IN-DEX 1.5 mcg/kg,

intranasal saline|Drug: Placebo - Saline

URL: https://ClinicalTrials.gov/show/NCT02773797

Study 13:

Title: A Comparison of Two Doses of Intranasal Dexmedetomidine for

Premedication in Children

Recruitment: Recruiting
Study Results: No Results Available Conditions: Anxiety, Separation
Interventions: Drug: Dexmedetomidine
URL: https://ClinicalTrials.gov/show/NCT02459509

Study 14:

Title: Pharmacokinetic Study of Dexmedetomidine After Intra-nasal Dosing in

Children

Study Results: No Results Conditions No Results Available

Conditions: Heart Disease

Interventions: Drug: Dexmedetomidine|Drug: Dexmedetomidine|Drug:

Dexmedetomidine

URL: https://ClinicalTrials.gov/show/NCT02836431

Study 15:

Title: Intranasal Dexmedetomidine for Procedural Pain Management in Elderly

Adults in Palliative Care

Recruitment: Not yet recruiting
Study Results: No Results Available
Conditions: Analgesia|Sedation|Anxiolysis

Interventions: Drug: Opioids|Drug: Dexmedetomidine|Drug: Placebo

URL: https://ClinicalTrials.gov/show/NCT03151863

Study 16:

Title: Premedication With Intranasal Dexmedetomidine or Midazolam for

Prevention of Emergence Agitation in Children
Recruitment: Not yet recruiting
Study Results: No Results Available
Conditions: Emergence Delirium

Conditions: Emergence Delirium
Interventions: Drug: Dexmedetomidine|Drug: Midazolam oral solution|Drug: Oral

saline|Drug: Nasal saline

URL: https://ClinicalTrials.gov/show/NCT03171740

Study 17:

Title: Intranasal Dexmedetomidine Premedication in Children

Recruitment: Completed Study Results: Has Results

Conditions: Preoperative Sedation

Interventions: Drug: Midazolam|Drug: Dexmedetomidine
URL: https://ClinicalTrials.gov/show/NCT02250703

Study 18:

Title: Intranasal Dexmedetomidine Sedation for Ophthalmic Examinations in

Children

Recruitment: Recruiting

Study Results: No Results Available

Conditions: Sniffs Drugs

Interventions: Drug: intranasal dexmedetomidine

URL: https://ClinicalTrials.gov/show/NCT02077712

Study 19:

Title: Sedation Using Intranasal Dexmedetomidine in Upper Gastrointestinal

Endoscopy

Recruitment: Completed

Study Results: No Results Available
Conditions: Gastrointestinal Disease
Interventions: Drug: Dexmedetomidine

URL: https://ClinicalTrials.gov/show/NCT01887184

Study 20:

Title: Comparison of Two Doses of Intranasal Dexmedetomidine as Premedication

in Children

Recruitment: Unknown status Study Results: No Results Available

Conditions: Patient Between 1-8 Years Old Undergoing Elective Surgery at Queen

Mary Hospital

Interventions: Drug: Dexmedetomidine

URL: https://ClinicalTrials.gov/show/NCT01065701

Study 21:

Title: Placebo-Controlled Evaluation of Intranasal Dexmedetomidine for

Postoperative Analgesia Following Bunionectomy Surgery

Recruitment: Completed
Study Results: Has Results
Conditions: Pain, Post-operative

Conditions: Pain, Post-operative
Interventions: Drug: Intranasal Dexmedetomidine|Drug: Intranasal Placebo

URL: https://ClinicalTrials.gov/show/NCT02284243

Study 22:

Title: A Trial Of Oral Chloral Hydrate Versus Intranasal Dexmedetomidine For

Sedated Abr Exams

Recruitment: Completed Study Results: Has Results Conditions: Sedation

Interventions: Drug: Chloral Hydrate|Drug: Dexmedetomidine|Other: Oral

placebo|Other: Intranasal placebo

URL: https://ClinicalTrials.gov/show/NCT01255904

Study 23:

Title: Placebo-Controlled Evaluation of Intranasal Dexmedetomidine for

Postoperative Analgesia Following Bunionectomy

Recruitment: Terminated
Study Results: Has Results
Conditions: Pain, Post-operative

Interventions: Drug: Intranasal Dexmedetomidine|Other: Intranasal Placebo

URL: https://ClinicalTrials.gov/show/NCT02169336

Study 24:

Title: Study Using Dexmedetomidine to Decreases Emergence Delirium in

Pediatric Patients

Recruitment: Unknown status
Study Results: No Results Available
Conditions: Otitis Media
Interventions: Drug: dexmedetomidine|Drug: saline
URL: https://ClinicalTrials.gov/show/NCT00778063

Study 25:

Dexmedetomidine in Children for Magnetic Resonance Imaging (MRI) Title:

Sedation

Recruitment:

Recruitment: Completed
Study Results: No Results Available
Conditions: Anesthesia
Interventions: Drug: Dexmedetomidine

URL: https://ClinicalTrials.gov/show/NCT02299232

Study 26: Title: Pharmacological Characteristics of Intranasally Given Dexmedetomidine in

Recruitment: Not yet recruiting
Study Results: No Results Available
Conditions: Procedural Sedation
Interventions: Device: Dexmedetomidine

URL: https://ClinicalTrials.gov/show/NCT02955732

Study 27:
Title: Dexmedetomidine Versus Fentanyl Following Pressure Equalization Tube
Placement

Recruitment: Completed Study Results: Has Results

Conditions: Chronic Otitis Media
Interventions: Drug: Dexmedetomidine|Drug: Fentanyl|Drug: Midazolam

https://ClinicalTrials.gov/show/NCT01188551 URL:

Study 28:

ED50 and ED95 of Intranasal Dexmedetomidine in Pediatric Patients

Undergoing Transthoracic Echocardiography Study

Recruitment: Recruiting

Study Results: No Results Available
Conditions: Patients for Transthoracic Echocardiography|Unknown Diagnosis
Interventions: Drug: intranasal dexmedetomidine

URL: https://ClinicalTrials.gov/show/NCT02780427

Study 29:

Intranasal Dexmedetomidine VS Oral Chloral Hydrate for Rescue Sedation

During Magnetic Resonance Imaging Recruitment: Completed

Study Results: No Results Available
Conditions: Administration Related Reaction|Failed Moderate Sedation During

Procedure|Chloral Hydrate Adverse Reaction

Interventions: Drug: chloral hydrate Group Drug: low dose dexmedetomidine

group|Drug: high dose dexmedetomidine group

https://ClinicalTrials.gov/show/NCT02239445 URL:

Study 30:

A Study to Assess the Analgesia and Sedation Using Intranasal

Dexmedetomidine in Third Molar Surgery Under Local Anaesthesia

Recruitment: Completed
Study Results: No Results Available
Conditions: Pain|Sedation
Interventions: Drug: Intranasal dexmedetomidine|Drug: Placebo
URL: https://ClinicalTrials.gov/show/NCT01132794

Study 31:

Title: The Effect of Age on the Median Effective Dose (ED50) of Intranasal Dexmedetomidine for Rescue Sedation Following Failed Sedation With Oral Chloral Hydrate

During Magnetic Resonance Imaging

Recruitment: Completed Study Results: No Results Available

Conditions: Aged|Drug|Dose-Response Relationship
Interventions: Drug: intranasal dexmedetomidine

URL: https://ClinicalTrials.gov/show/NCT02253199

### Australian New Zealand Clinical Trials Registry

### 4 Results

1.

The effects of ketamine on the quality of sedation of intranasal dexmedetomidine premedication in children undergoing elective tonsillectomy.

ACTRN12616001522404

Registered 20/11/2016

2.
Intranasal dexmedetomidine versus intranasal ketamine for prevention of emergence agitation after sevoflurane anesthesia in pediatric patients undergoing myringotomy: a randomized clinical trial.

ACTRN12616000921482

Registered

3

The Effect of Intranasal Dexmedetomidine Premedication on the Minimum Alveolar Concentration of Sevoflurane for tracheal intubation in children ACTRN12613000679785
Registered

28/06/2013

4

The Effect of Intranasal Dexmedetomidine Premedication on Reducing the Minimum Alveolar Concentration of Sevoflurane for the Insertion of Laryngeal Mask Airway in Children ACTRN12613000462785

Registered 25/04/2013

#### EU Clinical Trials Register

8 Results

EudraCT Number: 2016-002880-33 Sponsor Protocol Number: PINDEX Sponsor Name: University of Turku

Full Title: Bioavailability and pharmacokinetics of intranasal dexmedetomidine in

children

Start Date: 2016-10-28

Medical condition: Paediatric patients scheduled for minor procedures such as intra-articular

drug injections, hemia repair, bronchoscopy or magnetic resonance imaging.

Disease

Population Age: Children, Under 18 Gender: Male, Female Trial protocol: FI(Ongoing)

Link: https://www.clinicaltrialsregister.eu/ctrsearch/search?query=eudract\_number:2016-002880-33

EudraCT Number: 2016-002065-66 Sponsor Protocol Number: OY102016 Sponsor Name: Miikka Tervonen

Full Title: Intranasal dexmedetomidine sedation during intra-articular joint injections in

pediatric population

https://mc.manuscriptcentral.com/pediatrics

Start Date: 2016-11-07

Medical condition: All the patients from 1 year to 18 years of age who have been diagnosed by a pediatric rheumatologist to have a joint inflammation needing intra-articular corticosteroid

injection in 1 to 5 joints

Disease:

Population Age: Infants and toddlers, Children, Adolescents, Under 18, Adults

Gender: Male, Female Trial protocol: FI(Ongoing)

Link: https://www.clinicaltrialsregister.eu/ctrsearch/search?query=eudract\_number:2016-002065-66

EudraCT Number: 2016-001567-37 Sponsor Protocol Number: KUKIDEX-2

Sponsor Name: University Medical Center Groningen

Full Title: Efficacy of single dose intranasal dexmedetomidine for conscious sedation in

dental practice in dentophobic uncooperative patients with intellectual disability.

Start Date: 2016-11-24 Medical condition: dentophobia

intellectual disability

Disease:

Population Age: Adults
Gender: Male, Female
Trial protocol: NL(Ongoing)

Link: https://www.clinicaltrialsregister.eu/ctrsearch/search?query=eudract\_number:2016-001567-37

EudraCT Number: 2008-008324-33 Sponsor Protocol Number: 900, version 1.0

Sponsor Name: Sanna Vilo

Full Title: Bioavailability of dexmedetomidine after intranasal administration in healthy

subjects

Start Date: 2009-03-18

Medical condition: healthy volunteers

Disease:

Population Age: Adults, Elderly

Gender: Male

Trial protocol: FI(Completed)

Link: https://www.clinicaltrialsregister.eu/ctrsearch/search?query=eudract\_number:2008-008324-33

EudraCT Number: 2015-004587-11 Sponsor Protocol Number: KUKIDEX-1

Sponsor Name: University Medical Center Groningen

Full Title: Safety, tolerability and sedative properties of single dose intranasal

dexmedetomidine premedication in elderly subjects.

Start Date: 2016-01-08

Medical condition: Anxiety, preoperative

Disease:

Population Age: Elderly
Gender: Male, Female
Trial protocol: NL(Ongoing)

Link: https://www.clinicaltrialsregister.eu/ctrsearch/search?query=eudract\_number:2015-004587-11

EudraCT Number: 2017-000057-40 Sponsor Protocol Number: dex\_vs\_ket

Sponsor Name: Karolinska University Hospital

Full Title: A prospective randomized double-blind study Intranasal dexmedetomidine versus intranasal S-ketamine for children age 1 – 3 years for procedural sedation and analgesia

pediatric emergency departm... Start Date: 2017-06-12

Medical condition: sedation for emergency procedures

Disease:

Population Age: Infants and toddlers, Children, Under 18

Gender: Male, Female Trial protocol: SE(Ongoing)

Link: https://www.clinicaltrialsregister.eu/ctrsearch/search?query=eudract\_number:2017-000057-40

EudraCT Number: 2016-003773-17 Sponsor Protocol Number: dex version1

Sponsor Name: Karolinska University Hospital

Full Title: A prospective randomized open label study Intranasal dexmedetomidine versus inhaled nitrous oxide for children age 3 – 15 years for procedural sedation and analgesi

in pediatric emergency departme... Start Date: 2017-06-12

Medical condition: sedation for emergency procedures

Disease:

Population Age: Children, Adolescents, Under 18

Gender: Male, Female Trial protocol: SE(Ongoing)

Link: https://www.clinicaltrialsregister.eu/ctrsearch/search?query=eudract\_number:2016-003773-17

EudraCT Number: 2015-002102-37

Sponsor Name: Fundació Parc Taulí

Full Title: Open randomized clinical trial to compare the efficacy of hypotensive

anesthesia with clonidine or dexmedetomidine during endoscopic nasal surgery

Start Date: 2015-10-02

Medical condition: Nasosinusal endoscopic surgery in patients with chronic sinusitis and/or

nasal polyposis

Disease: Version: 18.0, SOC Term: 10021881 - Infections and infestations,

Classification Code: 10009137, Term: Chronic sinusitis, Level: PT

Disease: Version: 18.0, SOC Term: 10042613 - Surgical and medical procedures,

Classification Code: 10028755, Term: Nasal polypectomy, Level: PT

Population Age: Adults
Gender: Male, Female
Trial protocol: ES(Ongoing)

Link: https://www.clinicaltrialsregister.eu/ctrsearch/search?query=eudract\_number:2015-002102-37

#### WHO ICTRP 22 Results

| Recruitment<br>status | Prospective<br>Registration | <u>Main ID</u> | Public Title | <u>Date of</u><br><u>Registration</u> |
|---|---|---|---|---|
| Authorised | Yes | EUCTR2016-003773-<br>17-SE | Comparison of intranasally given drug dexmedetomidine with N2O (=laughing gas) for sedation for small procedures in children's emergency department. | 13/01/2017 |
| Authorised | Yes | EUCTR2017-000057-<br>40-SE | Comparison of intranasally given drug dexmedetomidine with intranasal S-keramine for sedation for small procedures in children's emergency department. | 13/01/2017 |
| Recruiting | Yes | ChiCTR-IIR-16010263 | Comparison of Rapid IV Bolus and Intranasal Adminstration of Dexmedetomidine for Treatment and | 2016-12-27 |

https://mc.manuscriptcentral.com/pediatrics

| | | | Prophylaxis of Emergence Agitation in Anesthetized Pediatric Patient | |
|---|---|---|---|---|
| Recruiting | Yes | NCT03069638 | Intranasal Dexmedetomidine Sedation During Intra- articular Joint Injections in Pediatric Population | 20/12/2016 |
| Recruiting | Yes | ChiCTR-OOC-<br>16009846 | Median Effective Dose of intranasal dexmedetomidine sedation for Pediatric transthoracic echocardiography between the children with and without history of cardiac operation: A Biased-Coin Up-and-Down Sequential Allocation Trial | 2016-11-13 |
| Recruiting | Yes | ChiCTR-OPC-<br>16009842 | Efficacy study of intranasal dexmedetomidine for pediatric sedation | 2016-11-13 |
| Recruiting | Yes | ChiCTR-IOR-<br>16009780 | Effects of intranasal dexmedetomidine combined with ketamine sedation for echocardiography in pediatric patients with congenitial heart disease | 2016-11-08 |
| Authorised | Yes | EUCTR2016-002065-<br>66-FI | Intranasal dexmedetomidine sedation during intra- articular joint injections in pediatric population | 02/11/2016 |

https://mc.manuscriptcentral.com/pediatrics

| Authorised | Yes | EUCTR2016-002880-<br>33-FI | Pharmacological<br>characteristics of<br>intranasally given<br>dexmedetomidine in<br>paediatric patients | 17/10/2016 |
|---|---|---|---|---|
| Authorised | Yes | EUCTR2016-001567-<br>37-NL | Efficacy of dexmedetomidine for conscious sedation during dental treatement of uncooperative patients with intellectual disability and fear of dentists. | 20/07/2016 |
| Recruiting | Yes | NCT02780427 | ED50 and ED95 of<br>Intranasal Dexmedetomidine in Pediatric Patients Undergoing Transthoracic Echocardiography Study | 12/05/2016 |
| Recruiting | Yes | IRCT201601281882N7 | Premedication effect of intranasal midazolam and dexmedetomidine on children behavior | 2016-03-13 |
| Recruiting | Yes | ChiCTR-IOR-<br>16008076 | Evaluation of Efficacy<br>and Safety of Intranasal<br>Dexmedetomidine<br>Premedication for<br>Hypertension Patients | 2016-03-09 |
| Recruiting | Yes | NCT02836431 | Pharmacokinetic Study of<br>Dexmedetomidine After<br>Intra-nasal Dosing in<br>Children | 08/01/2016 |
| Authorised | Yes | EUCTR2015-004587-<br>11-NL | Is dexmedetomidine a safe medicine to calm elderly patients when they are waiting for an operation? | 17/12/2015 |

| Recruiting | Yes | NCT02459509 | A Comparison of Two Doses of Intranasal Dexmedetomidine for Premedication in Children | 20/05/2015 |
|---|---|---|---|---|
| Recruiting | Yes | ChiCTR-TRC-<br>14004886 | A randomized, double-<br>blind assessment of the<br>sedative and analgesic<br>effects of intranasal<br>dexmedetomidine in nasal<br>endoscopic surgery cases | 2014-07-02 |
| Recruiting | Yes | NCT02108171 | Intranasal<br>Dexmedetomidine<br>Premedication | 30/03/2014 |
| Recruiting | Yes | NCT02077712 | Intranasal Dexmedetomidine Sedation for Ophthalmic Examinations in Children | 27/02/2014 |
| Recruiting | Yes | NCT01900405 | Intranasal Dexmedetomidine Sedation for Pediatric CT Imaging | 09/07/2013 |
| Recruiting | No | NCT01065701 | Comparison of Two Doses of Intranasal Dexmedetomidine as Premedication in Children | 07/02/2010 |
| Recruiting | Yes | NCT00778063 | Study Using Dexmedetomidine to Decreases Emergence Delirium in Pediatric Patients | 21/10/2008 |

#### Conference Abstracts

Association of Anaesthetists of Great Britain and Ireland Annual Congress (2012-2016) American Society for Pediatric Anesthesia Annual Meeting (2013-2016) Canadian Anesthesiologists' Society Annual Meeting (2012-2015) The Congress of the European Pain Federation (2013-2015)

European Society of Intensive Care Medicine (2012-2016)
European Society of Anaesthesiology (2012-2016)
European Society of Regional Anaesthesia (2012-2016)
Canadian Association of Emergency Physicians (2012-2017)
Society of Academic Emergency Medicine (2012-2016)
Australasian College for Emergency Medicine (2012-2016)
International Federation on Emergency Medicine (2012)
European Society of Emergency Medicine (2013-2016)
Canadian Paediatric Society (2014-2016)

List word counts below (do not paste the text here). Please see the Decision Letter Attachment for allowances as they pertain to your manuscript type.

```
# of words in Abstract: 250 (250 words allowed)
```

- # of words in Manuscript Body: 3685 (3000 allowed for Regular Articles/Quality Reports; 4000 Reviews/Special Articles; 800 Commentaries; 1200 Perspectives)
- # of characters in Main Title: 83 characters (97 characters allowed, including spaces)
- # of characters in Short Title: 50 (55 characters allowed, including spaces)
- # of words in "Table of Contents Summary": 19 (25 words allowed; this section appears in all articles with abstracts)
- # of words in "What's Known on this Subject": 40 (40 words allowed; this section appears in Regular Articles only)
- # of words in "What this Study Adds": 40 (40 words allowed; this section appears in Regular Articles only)

#### 2019-1623.R2 - Intranasal dexmedetomidine for procedural distress in children: a systematic review -- by Poonai et al.

| EDITOR/REVIEWER COMMENTS | AUTHOR'S RESPONSE | REFERENCE PAGE | CHANGE |
|---|---|---|---|
| Paste each of the editor and reviewer | Paste your answer to the editor and reviewer queries here. | State where* the | APPROVED? |
| queries here. | If you alter your manuscript to address this query, you MUST paste the relevant altered | change now | FOR |
| | text here – verbatim as it appears in the manuscript. | appears in your | EDITORIAL USE |
| | | newly revised | ONLY |
| | | manuscript. | |
| EXAMPLE: Reviewer 1's comment | EXAMPLE: A brief response to this reviewer's comment. | EXAMPLE 1: | |
| | | Page 7, lines 10- | |
| | The text now states: "insert relevant changed text here" | 22 | |
| | | EXAMPLE 2: | |
| | | No change | |
| Please consider rewriting the abstract | Thank you. The following changes to the abstract results have been made with respect | Abstract | |
| results to make it a bit less confusing | to wording. | | |
| | The terms "favorable", "neutral", and "unfavorable" were replaced with "superior", | | |
| | "equivalent", and "inferior" to improve readability and general comprehension. | | |
| Change the short title (both in your paper | The short title has been changed. | Title | |
| and in online Step 1) to: Intranasal | | | |
| dexmedetomidine for procedural distress | | | |
| The sedation instruments used by various | We initially removed this part of the text to reduce the word count. We have added this | Page 9, lines 256- | |
| studies has been removed from the current | back in as per your recommendation. | 259 | |
| version. It was there is the initial | | | |
| submission. I am wondering if there a | A validated sedation instrument was used in ten trials (25-27, 29-34, 36) and included | | |
| specific reason the authors removed it from | the Observer's Assessment of Alertness/Sedation, Modified Observer's Assessment of | | |
| the revised version. If there is no reason it | Alertness/Sedation Scale, Ramsay Sedation Scale, and the University of Michigan | | |
| may be better to add it back. | Sedation Scale (Table 1). | | |
| | 7 | | |
| | I | I | |

| Line 262: The authors may have | We have made this correction. | Page 9-10, lines |
|---|---|---|
| inadvertently omitted "participants"—"The | | 263-264 |
| proportion with adequate sedation was | The proportion of participants with adequate sedation was 33/41 (80.4%) for IND plus | |
| 33/41 (80.4%) participants (?). " Otherwise | oral ketamine | |
| it is a little confusing as to what it means. It | | |
| is present in the rest of the manuscript. | | |
| The authors have reported the overall | Thank you for this comment. The revised (last submitted) version reports adverse events | Page 12, lines |
| adverse events. Would they be able to | per interventions which are groups as follows: IND, IND + another sedation, and non-IND | 322-327 |
| comment if the adverse events- particularly | comparator. Bradycardia and hypotension are listed first. Inferential statistics were not | |
| bradycardia and hypo/hypertension was | performed because the meta-analysis was deconstructed for all outcomes including | |
| greater with IND (or similar). I think it was<br>reported in the initial submission. | adverse events. The section reads: | |
| | Across the remaining 18 trials, the most common adverse events of IND, IND plus | |
| | another sedative, or non-IND comparator were bradycardia [32/1484 (2.2%), 0/41 (0%), | |
| | and 6/595 (1%), respectively], hypotension [18/1484 (1.2%), 0/41(0%), and 9/595 (1.5%), | |
| | respectively], oxygen desaturation [7/1484 (0.5%), 0/41 (0%), and 12/595 (2%), | |
| | respectively], and vomiting [6/1484 (0.4%), 3/41 (7.3%), and 47/595 (7.9%), | |
| | respectively]. | |
| 2nd para: The NICE guidelines are from | This is a very important point and we thank you for raising it. The section has been | Page 13-14, lines |
| 2010. Chloral hydrate is no longer available | revised to read: | 354-355 |
| in the United States. | | |
| https://medlineplus.gov/druginfo/meds/a6 | In fact, chloral hydrate is recommended by the National Institute for Health and Care | |
| 82201.html | Excellence (NICE) 2010 guideline for moderate sedation for painless procedures in | |
| | children (44). While chloral hydrate is no longer approved by the United States Food and | |
| I think it is completely acceptable that this | Drug Administration, it may still be used in other countries. | |
| review looked at chloral hydrate as one of | | |
| the comparators. It may still be used in | | |
| other countries. However, it is important<br>that the above information that it is not | | |
| approved by the FDA should be included - | | |
| since this article will be reaching | | |
| pediatricians in the US as well. | | |
| pediatricians in the US as well. | | |

#### Instructions:

Please use this table format to answer the questions posed by the editors and reviewers of your paper. Copy and paste the editor/reviewer's question in the "Comments" column and your answer to that question in the corresponding "Response" column. Be sure to ALSO paste the corrected text along with your response. For minor copyediting changes such as spelling and grammar corrections, you may simply state that the error was corrected, without pasting the altered text.

\* Use the page/line numbers from your revised .doc, .rtf, or .txt file; do not use the page/line numbers from the submission system's auto-generated PDF.

For clarity, use one row per question. Make sure to list the page and line reference where your change can be found. If no change was made, please make sure to note

### **Appendix B Pediatric Sedation State Scale (PSSS)**

#### TABLE 2 PSSS

| State | Behavior |
|---|---|
| 5 | Patient is moving (purposefully or nonpurposefully) in a manner that impedes the proceduralist and requires forceful immobilization. This includes crying or shouting during the procedure, but vocalization is not required. Score is based on movement. |
| 4 | Moving during the procedure (awake or sedated) that requires gentle immobilization for positioning. May verbalize some discomfort or stress, but there is no crying or shouting that expresses stress or objection. |
| 3 | Expression of pain or anxiety on face (may verbalize discomfort), but not moving or impeding completion of the procedure. May require help positioning (as with a lumbar puncture) but does not require restraint to stop movement during the procedure. |
| 2 | Quiet (asleep or awake), not moving during procedure, and no frown (or brow furrow) indicating pain or anxiety. No verbalization of any complaint. |
| 1 | Deeply asleep with normal vital signs, but requiring airway intervention and/or assistance (eg. central or obstructive apnea, etc). |
| 0 | Sedation associated with abnormal physiologic parameters that require acute intervention (ie, oxygen saturation <90%, blood pressure is 30% lower than baseline, bradycardia receiving therapy). |

### Appendix C

The Council for International Organizations of Medical Sciences (CIOMS)

| | | | | | | | | | | | CIOMS FORM |
|---|---|---|---|---|---|---|---|---|---|---|---|
| SUSPECT ADV | ERSE REACTI | ION REPORT | т | | | | | | | | |
| SOSPECT ADV | ENSE NEACT | ION INEL OIL | ' | | | | Т | П | | Т | |
| I. REACTION INFORMATION 1. PATIENT INITIALS 1a. COUNTRY 2. DATE OF BIRTH 2a. AGE 3. SEX 4-6 REACTION ONSET | | | | | | | | | | | |
| 1. PATIENT INITIALS (first, last) | 1a. COUNTRY | 2. DATE OF E | | Years | 3. SEX | Day | _ | | _ | _ | 8-12 CHECK ALL APPROPRIATE TO ADVERSE REACTION |
| 7 + 13 DESCRIBE F | REACTION(S) (inc | cluding relevan | t tests | /lab data | a) | | | | | | □ PATIENT DIED |
| | | | | | | | | ☐ INVOLVED OR PROLONGED INPATIENT HOSPITALISATION | | | |
| | | | | | | | | | | | INVOLVED PERSISTENCE OR SIGNIFICANT DISABILITY OR INCAPACITY |
| | | | | | | | | □ LIFE<br>THREATENING | | | |
| | II. SUSPECT DRUG(S) INFORMATION | | | | | | | | | | |
| 14. SUSPECT DRUG(S) (include generic name) | | | | | | | | 20 DID REACTION ABATE AFTER STOPPING DRUG? YES NO NA | | | |
| 15. DAILY DOSE(S) | | | | 16. RO | JTE(S) O | F ADM | ΛIN | STRA | TION | | 21. DID REACTION<br>REAPPEAR<br>AFTER REINTRO- |
| 17. INDICATION(S) FO | OR USE | | | | | | | | | | DUCTION? |
| 18. THERAPY DATES | (from/to) | | | 19. TH | IERAPY | DURA | TI | NC | | | |
| | III. CC | ONCOMITAN | NT DF | RUG(S) | AND | HIST | ΓΟΙ | RY | | | |
| 22. CONCOMITANT D | RUG(S) AND DA | TES OF ADMI | NISTRA | ATION ( | exclude | those | us | ed to | trea | at re | eaction) |
| 23. OTHER RELEVANT | HISTORY (e.g. | diagnostics, al | lergics | , pregna | ncy with | h last | me | onth | of pe | erioc | i, etc.) |
| | IV | . MANUFAC | TUR | FR INF | ORMA | TION | N. | | | | |
| 24a. NAME AND ADD | | | | , , ,,,,, | | | • | | | | |
| | 24b. MF | R CONTROL N | NO. | | | | | | | | |
| 24c. DATE RECEIVED<br>BY MANUFACTURE | RER □ STU | PORT SOURCE<br>DY DITERAT | TURE | | | | | | | | |
| DATE OF THIS REPORT | | PORT TYPE | WUP | | | | | | | | |

#### Appendix D

#### Post-Hospital Behavior Questionnaire (PHBQ)- Follow up between 24 to 48 hours after discharge (Hilly J, 2015)

| 1 Does | vour child | make a fuse | ahout going | to bed at night? |
|---------|-------------|-------------|-------------|------------------|
| I. DUCS | your cilliu | make a rus. | about going | to bed at might: |

| Much less than before (1) | Less than before (2) | Same as before (3) | More than before (4) | Much more than before (5) |
|---|---|---|---|---|
| 2. Does your child make a fu | uss about eating? | | | |

| Much less than before (1) | Less than before (2) | Same as before (3) | More than before (4) | Much more than before (5) |
|---|---|---|---|---|

3. Does your child spend time just sitting or lying and doing nothing?

| Much less than before (1) Less tha | n before (2) Sam | me as before (3) | More than before (4) | Much more than before (5) |
|---|---|---|---|---|
|---|---|---|---|---|

4. Does your child need a pacifier?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

5. Does your child seem to be afraid of leaving the house with you?

6. Is your child uninterested in what goes on around him (or her)?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

7. Does your child wet the bed at night?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

8. Does your child bite his (or her) finger nails?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

9. Does your child get upset when you leave him (or her) alone for a few minutes?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

10. Does your child need a lot of help doing things?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

11. Is it difficult to get your child interested in doing things (like playing games with toys/video games)?

12. Does your child seem to avoid or be afraid of new things?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

13. Does your child have difficulty making up his (or her) mind?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

14. Does your child have temper tantrums?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

15. Is it difficult to get your child to talk to you?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

16. Does your child seem to get upset when someone mentions doctors or hospitals?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

17. Does your child follow you everywhere around the house?

| 18. Does your child spend time trying to get or hold your attention? |
|----------------------------------------------------------------------|

| Much less than before (1) | Less than before (2) | Same as before (3) | More than before (4) | Much more than before (5) |
|---|---|---|---|---|

| Much less than before (1) | Less than before (2) | Same as before (3) | More than before (4) | Much more than before (5) |
|---|---|---|---|---|

20. Does your child have bad dreams at night or wake up and cry?

| Much less than before (1) | Less than before (2) | Same as before (3) | More than before (4) | Much more than before (5) |
|---|---|---|---|---|

21. Does your child have irregular bowel movements?

| Much less than before (1) | Less than before (2) | Same as before (3) | More than before (4) | Much more than before (5) |
|---|---|---|---|---|

22. Does your child have trouble getting to sleep at night?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

23. Does your child seem to be shy around strangers?

24. Does your child have a poor appetite?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

25. Does your child tend to disobey you?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

26. Does your child break toys or other objects?

Much less than before (1) Less than before (2) Same as before (3) More than before (4) Much more than before (5)

27. Does your child suck his (or her) fingers or thumbs?

**Appendix E** 

PRODUCT MONOGRAPH

PRECEDEX®

Dexmedetomidine Hydrochloride for Injection 100 mcg/mL dexmedetomidine (as dexmedetomidine hydrochloride) (Concentrate, 2 mL vial)

Dexmedetomidine Hydrochloride Injection 4 mcg/mL dexmedetomidine (as dexmedetomidine hydrochloride) (Ready to use, 20 mL, 50 mL and 100 mL vials)

Alpha2-adrenergic agonist

Pfizer Canada Inc. 17300 Trans-Canada Highway Kirkland, Québec H9J 2M5

Submission Control No.: 213361

Date of Revision: March 6, 2018

#### **Table of Contents**

| PART I: HEALTH PROFESSIONAL INFORMATION | 3 |
|-----------------------------------------------------------|----|
| SUMMARY PRODUCT INFORMATION | 3 |
| INDICATIONS AND CLINICAL USE | 3 |
| CONTRAINDICATIONS | 4 |
| WARNINGS AND PRECAUTIONS | 4 |
| ADVERSE REACTIONS | 7 |
| DRUG INTERACTIONS | 12 |
| DOSAGE AND ADMINISTRATION | |
| OVERDOSAGE | 15 |
| ACTION AND CLINICAL PHARMACOLOGY | 15 |
| STORAGE AND STABILITY | 19 |
| SPECIAL HANDLING INSTRUCTION | 20 |
| DOSAGE FORMS, COMPOSITION AND PACKAGING | 22 |
| PART II: SCIENTIFIC INFORMATIONPHARMACEUTICAL INFORMATION | 23 |
| CLINICAL TRIALS | |
| DETAILED PHARMACOLOGY | |
| TOXICOLOGY | |
| REFERENCES | 30 |
| PART III: CONSUMER INFORMATION | 32 |



#### Dexmedetomidine Hydrochloride for Injection Dexmedetomidine Hydrochloride Injection

#### PART I: HEALTH PROFESSIONAL INFORMATION

#### SUMMARY PRODUCT INFORMATION

| Route of<br>Administration | Dosage Form / Strength | All Nonmedicinal<br>Ingredients |
|---|---|---|
| Intravenous | Parenteral injection,100 mcg/mL in a 2 mL vial (Concentrate) | Sodium Chloride and Water |
| infusion | Parenteral injection,4 mcg/mL in 20 mL,<br>50 mL and 100 mL vials (Ready to Use) | for Injection |

#### INDICATIONS AND CLINICAL USE

Precedex<sup>®</sup> (Dexmedetomidine Hydrochloride for Injection and Dexmedetomidine Injection) is indicated for:

#### • Intensive Care Unit Sedation

Precedex<sup>®</sup> is indicated for sedation of initially intubated and mechanically ventilated patients during treatment in an intensive care setting by continuous intravenous infusion. The Precedex<sup>®</sup> infusion should not generally exceed 24 hours.

Precedex<sup>®</sup> has been continuously infused in mechanically ventilated patients prior to extubation, during extubation, and post-extubation. It is not necessary to discontinue Precedex<sup>®</sup> prior to extubation.

#### Conscious Sedation

Precedex<sup>®</sup> is indicated for sedation of non-intubated patients prior to and/or during surgical and other procedures by continuous intravenous infusion for the following procedures:

- Monitored Anesthesia Care (MAC) with an adequate nerve block and/or local infiltration;
- Awake Fiberoptic Intubation (AFI) with adequate topical preparation of the upper airway with local lidocaine formulations.

Due to insufficient safety and efficacy data, Precedex<sup>®</sup> is not recommended for use in procedures other than the two listed above.

| The picture can't be displayed. |
|---------------------------------|

| The picture can't be displayed. |
|---------------------------------|
| The become over 60 embedden |

| The picture can't be displayed. | $\neg$ |
|---------------------------------|--------|
| <u>-</u> | |
| L | |

| The picture can't be displayed. |
|---------------------------------|
| I |

| The picture can't be displayed. |
|---|
| - Inches of the property of th |

| The picture can't be displayed. |
|---|
| The present sent to the supplying the supply |

| ▼ The picture can't be displayed. |
|-----------------------------------|

| Study: Intranasal dexmedetomidine for lacera | tion repair in children: a dose-finding study |
|---|---|
| Protocol: Dose Finding Study | Version 3.2 – August 12, 2019 |

| The picture can't be displayed. | |
|---------------------------------|------|
| | - 00 |

| Respiratory System Disorders | Apnea, bronchospasm, dyspnea, hypercapnia, hypoventilation, |
|---|---|
| | hypoxia, pulmonary congestion |
| Skin and Appendages Disorders | Increased sweating |
| Vascular disorders | Hemorrhage |
| Vision Disorders | Photopsia, abnormal vision |

#### DRUG INTERACTIONS

#### **Drug-Drug Interactions**

#### Anesthetics, sedatives, hypnotics, opioids

Co-administration of Precedex® with anesthetics, sedatives, hypnotics, and opioids is likely to lead to an enhancement of effects. Specific studies have confirmed enhanced effects with sevoflurane, isoflurane, propofol, alfentanil, and midazolam. No pharmacokinetic interactions between Precedex® and isoflurane, propofol, alfentanil and midazolam have been demonstrated. However, due to possible pharmacodynamic interactions, when co-administered with Precedex®, a reduction in dosage of Precedex® or the concomitant anesthetic, sedative, hypnotic or opioid may be required.

#### Neuromuscular Blockers

In one study of 10 healthy adult volunteers, administration of Precedex<sup>®</sup> for 45 minutes at a plasma concentration of 1 (one) ng/mL resulted in no clinically meaningful increases in the magnitude of neuromuscular blockade associated with rocuronium administration.

#### Drugs with cardiovascular activities

Precedex® is known to be associated with hypotension and bradycardia, especially during its initial use. However, it may also be associated with a transient or paradoxical hypertension which may occur during the initial use and maintenance use. Concomitant medications acting on the cardiovascular system should be reviewed, in addition to reducing the dexmedetomidine dose and/or using a vasodilator.

#### Cytochrome P-450

*In vitro* studies in human liver microsomes demonstrated no evidence of cytochrome P450 mediated drug interactions that are likely to be of clinical relevance.

#### DOSAGE AND ADMINISTRATION

#### **Dosing Considerations**

- Precedex<sup>®</sup> should be used only in facilities adequately staffed and equipped for anesthesia, resuscitation, and cardiovascular monitoring.
- Precedex<sup>®</sup> should not be generally used for duration longer than 24 hours. Its continued use beyond 24 hours should be determined based on careful assessment of the patient's conditions.
- Precedex<sup>®</sup> should be administered using a controlled infusion device with adequate precision.

| The picture can't be displayed. |
|---------------------------------|

| The picture can't be displayed. |
|---------------------------------|
| _ |
| L |

| The picture can't be displayed. |
|---------------------------------|

| Study: Intranasal dexmedetomidine for lace | ration repair in children: a dose-finding study |
|---|---|
| Protocol: Dose Finding Study | Version 3.2 – August 12, 2019 |

| X The picture can't be displayed. |
|-----------------------------------|

| The picture can't be displayed. |
|---------------------------------|
| • |

| The picture can't be displayed. |
|---------------------------------|
| - |

| The picture can't be displayed. | |
|---------------------------------|-----|
| | 107 |
| The picture can't be displayed. | |
|---------------------------------|--|

| The picture can't be displayed. |
|---------------------------------|

| The sides and he distributed |
|---------------------------------|
| The picture can't be displayed. |

| [n | _ |
|---------------------------------|---|
| The picture can't be displayed. | |
| I . | |

| The picture can't be displayed. |
|---------------------------------|
| <u></u> |
| • |

| The picture con't be displayed. |
|---------------------------------|

| ▼ The picture can't be displayed. |
|-----------------------------------|

Dexmedetomidine given intravenously is devoid of clear CNS activity up to 0.001 mg/kg in mice and rats; at higher doses ( $\geq 0.003 \text{ mg/kg}$ ), dexmedetomidine induced clear CNS depressant effects.

#### **Pharmacokinetics**

In beagle dogs, dexmedetomidine was rapidly eliminated following a 50 mcg/kg IV dose with a mean apparent  $t_{1/2}$  of 0.68 hour; plasma elimination  $t_{1/2}$  was slightly longer following intramuscular (IM) dosing.

Rats administered an intravenous 20 mcg/kg dose of [<sup>3</sup>H]dexmedetomidine showed drugrelated radioactivity widely distributed throughout the body, with the highest mean concentrations in blood, plasma, and selected tissues occurring from 0.25 to 12 hours postdose.

[<sup>3</sup>H]dexmedetomidine was extensively metabolized by rats. Less than 1% of the dose was excreted in the urine as the parent drug. Major urinary metabolites included the COOH, OH, G-OH, SO<sub>3</sub>OH, M-2, and M-5 metabolites. Levels of the SO<sub>3</sub>OH metabolite were greater in female urine than in male urine. Fecal patterns generally resembled those found in urine.

The metabolism of [³H]dexmedetomidine in beagle dogs was similar to that observed in rats. Biliary excretion of [³H]dexmedetomidine following IV and SC administration was studied in rats with an implanted bile-duct cannula; an average of 51.6% and 45.4% of the radioactive dose was recovered in rat bile 24 hours after IV and SC administration, respectively. Major biliary metabolites were the glucuronide of a hydroxylated metabolite (G-OH) and an unidentified conjugate, M-2. Unidentified metabolites represented 12% to 18% of the dose.

Lacteal excretion, tissue distribution, and placental transfer of radioactivity were studied in rats following administration of a 0.015 mg/kg SC dose of [³H]dexmedetomidine. Radioactivity was distributed in maternal tissues and crossed the placenta to distribute in fetal tissues. Drug-related radioactivity was detected in the milk of dams at 0.5 hours and reached a maximum mean concentration at 4 hours. Thereafter, levels of radioactivity in milk decreased to non-detectable levels at 72 hours. The milk:plasma concentration ratio was less than 1 at all collection time points, indicating that radioactivity did not accumulate in the milk.

#### TOXICOLOGY

#### Acute Toxicity

The highest non-lethal dose by intravenous injects was 1000 mcg/kg in mice, rats and dogs in both sexes.

In a rat neurotoxicity study, Day 7 postnatal rat pups subcutaneously injected with Precedex<sup>®</sup> (3 mcg/kg or 10 mcg/kg or 30 mcg/kg), did not produce significant degeneration in the limbic thalamic nuclei and limbic cortical regions compared to ketamine (20 mg/kg), which resulted in significant neuronal cell death and degeneration. This was determined by histological staining

(silver, Fluoro-Jade B, and Caspase-3) to detect neuroapoptosis and neurodegeneration in postnatal rat pup brains.

#### Long-Term Toxicology

A two-week IV infusion study in adult dogs was performed to investigate the potential effect of dexmedetomidine on toxicologic, pathologic, and hormone secretion parameters. Dexmedetomidine at 50 or 100 mcg/kg/day was well-tolerated, with treatment-related effects (sedation, hypothermia (\$\pm\$ 3-4°C)) reversed by the end of the recovery period. Dexmedetomidine increased cortisol secretion, decreased LH secretion in males, decreased TSH secretion, and at the 100 mcg/kg/day dose level, decreased ACTH-stimulated cortisol secretion.

Rats receiving dexmedetomidine by IV administration for four weeks at doses up to 160 mcg/kg/day showed sedation and piloerection occurring at all doses, with exophthalmos observed only at the highest dose. No deaths occurred. Based on the drug-related small decreases in thymus and body weights at 160 mcg/kg/day, the no-toxic-effect-dose (NTED) of dexmedetomidine was determined to be 40 mcg/kg/day.

#### Carcinogenicity

Animal carcinogenicity studies have not been performed with dexmedetomidine.

#### Genotoxicity

Dexmedetomidine was not found to be mutagenic in the Ames *Salmonella* and *E. coli* assays, L5178/tk<sup>+/-</sup> mouse lymphoma assay, in vitro human lymphocyte cytogenics assays, and in vivo mouse micronucleus assays. No structural or numerical chromosome aberrations were noted in the presence or absence of metabolic activation. Dexmedetomidine did not demonstrate clastogenic activity.

#### Reproductive Toxicology

Reproductive and developmental toxicity studies were performed with dexmedetomidine in rats and rabbits.

A fertility study (Segment I) in rats at doses up to 54 mcg/kg/day administered subcutaneously showed that the No-Observed-Adverse-Effect Level (NOAEL) for F0 males and females was 54 mcg/kg/day for fertility indices and 6 mcg/kg/day for systemic toxicity. The NOAEL for F1 development was considered to be at 6 mcg/kg/day.

In a prenatal monkey neurotoxicity study, infusion of Precedex to pregnant monkeys at doses up to 30 mcg/kg/hr (10X Human Equivalent Dose) for 12 hours did not induce neuroapoptosis in fetal monkey brains compared to controls. In the same study, infusion of ketamine at 20-50 mg/kg/hr for 12 hours to mothers resulted in significant neuroapoptosis in fetal monkey brains. This was determined by immunohistochemical staining for activated caspase 3 and TUNEL in fetal monkey brains.

Teratogenic effects were not observed following administration of dexmedetomidine at subcutaneous doses up to 200 mcg/kg in rats from day 5 to day 16 of gestation and intravenous doses up to 96 mcg/kg in rabbits from day 6 to day 18 of gestation. The dose in rats is

approximately 2 times the maximum recommended human intravenous dose on a mcg/m² basis. The exposure in rabbits is approximately equal to that in humans at the maximum recommended intravenous dose based on plasma area-under-the-curve values. However, fetal toxicity, as evidenced by increased post-implantation losses and reduced live pups, was observed in rats at subcutaneous dose of 200 mcg/kg. The no-effect dose was 20 mcg/kg (less than the maximum recommended human intravenous dose on a mcg/m² basis). In another reproductive study when dexmedetomidine was administered subcutaneously to pregnant rats from gestation day 16 through nursing, it caused lower pup weights at 8 and 32 mcg/kg as well as fetal and embryocidal toxicity of second generation offspring at a dose of 32 mcg/kg (less than the maximum recommended human intravenous dose on a mcg/m² basis). Dexmedetomidine also produced delayed motor development in pups at a dose of 32 mcg/kg (less than the maximum recommended human intravenous dose on a mcg/m² basis). No such effects were observed at a dose of 2 mcg/kg (less than the maximum recommended intravenous dose on a mcg/m² basis). Placental transfer of dexmedetomidine was observed when radiolabeled dexmedetomidine was administered subcutaneously to pregnant rats.

In rabbits, the influence of dexmedetomidine on teratogenicity (Segment II) after IV administration in doses up to 96 mcg/kg/day was investigated. The NOAEL was 96 mcg/kg/day for maternal toxicity and 96 mcg/kg/day for F1 development. No higher dose was feasible. No teratogenicity was observed in any dose level tested.

Prenatal and postnatal development (Segment III study) was examined in rats at doses up to 32 mcg/kg/day administered subcutaneously. The NOAEL was 8 mcg/kg/day for maternal toxicity and 2 mcg/kg/day for F1 development.

#### **Local Tolerance Studies**

A solution of dexmedetomidine was shown to be mildly irritating in rats when injected intramuscularly.

#### REFERENCES

- Aantaa R, Kallio A, Virtanen R. Dexmedetomidine, a novel α-2-adrenergic agonist. A review of its pharmacodynamic characteristics. Drugs of the Future. 1993;18(1):49-56.
- Candiotti, K et al. Monitored Anesthesia Care with Dexmedetomidine: A Prospective, Randomized, Double-Blind, Multicenter Trial. Ambulatory Anesthesia. 2010: Vol. 110, No. 1 pp. 47-56.
- Chrysostomou, C et al. A Phase II/III, Multicenter, Safety, Efficacy, and Pharmacokinetic Study of Dexmedetomidine in Preterm and Term Neonates. *J Pediatr* 2014 Feb; 164(2): 276-82.
- De Jonghe B, Cook D, Appere-De-Vecchi C, et al. Using and understanding sedation scoring systems: a systemic review. *Intensive Care Med.* 2000;26:275-85.
- DeWolf AM, Fragen RJ, Avram MJ, et al. The pharmacokinetics of dexmedetomidine in volunteers with severe renal impairment. Anesth Analg. 2001;93:1205-1209.
- Dyck JB, Shafer SL. Dexmedetomidine pharmacokinetics and pharmacodynamics. *Anaesth Pharm Rev.* 1993;1(3):238-245.
- Ebert TJ, Hall JE, Barney JA, et al. The effects of increasing plasma concentrations of dexmedetomidine in humans. *Anesthesiology*. 2000;93:382-394.
- 8. Fraser GL, et al. Evaluation of agitation in ICU patients: incidence, severity and treatment in the young versus the elderly. *Pharmacotherapy*. 2000;20:75-82.
- Herr DL, Sum-Ping STJ, England M. ICU sedation after coronary artery bypass graft surgery: dexmedetomidine-based versus propofol-based sedation regimens. J Cardiothorac Vasc Anesth. 2003;17(5):576-584.
- Jakob SM, et al. Dexmedetomidine vs Midazolam or Propofol for Sedation During Prolonged Mechanical Ventilation Two Randomized Controlled Trials. *JAMA* 2012;307 (11): 1151-1160
- Kamibayashi T, Maze M. Clinical uses of alpha-2-adrenergic agonists. *Anesthesiology* 2000;93:1345-9.
- Martin E, Ramsay G, et al. The Role of the alpha-2 Adrenoreceptor Agonist Dexmedetomidine in Postsurgical Sedation in the Intensive Care Unit. *Journal of Intensive Care Medicine*. 2003 Vol. 18 No. 7; 29-41

#### PART III: CONSUMER INFORMATION

<sup>®</sup>Precedex<sup>®</sup>

Dexmedetomidine Hydrochloride for Injection Dexmedetomidine Hydrochloride Injection

This leaflet is part III of a three-part "Product Monograph" published when Precedex® was approved for sale in Canada and is designed specifically for Consumers. This leaflet is a summary and will not tell you everything about Precedex®. Contact your doctor or pharmacist if you have any questions about the drug.

#### ABOUT THIS MEDICATION

#### What the medication is used for:

Precedex® is used in adults:

- for continuous sedation (to keep you calm) after you arrive at the intensive care unit after your surgery under a general anesthesia
- for sedation when you receive certain surgical procedures under a local anesthesia or nerve block or when you receiving a breathing tube while awake

#### What it does:

Precedex acts by activating a part of the brain which helps keep you calm.

#### When it should not be used:

You should not be given Precedex® if you:

 are allergic to dexmedetomidine hydrochloride or to any non-medicinal ingredient in the formulation.

#### What the medicinal ingredient is:

dexmedetomidine hydrochloride.

#### What the nonmedicinal ingredients are:

sodium chloride and water for injection. Precedex is preservative-free and contains no additives or other chemicals.

#### What dosage forms it comes in:

Precedex is available as:

- A solution containing 100 micrograms/mL of dexmedetomidine that will be further diluted into saline and given to you by intravenous infusion. The Precedex® concentrate solution is available in a 2 mL glass vial.
- A solution containing 4 micrograms/mL of dexmedetomidine that is ready to use. No dilution is required. The Precedex<sup>®</sup> ready to use solution is available in 20 mL, 50 mL and 100 mL glass vials.

#### WARNINGS AND PRECAUTIONS

Precedex<sup>®</sup> should only be administered by healthcare professionals skilled in the management of patients in the intensive care unit or operating room setting.

### BEFORE you are given Precedex<sup>®</sup> talk to your doctor or nurse if you:

- have heart problems, including chronic high blood pressure
- have diabetes mellitus
- have liver problems
- have severe kidney problems
- · are taking any other medicines
- are dehydrated or suffer from excessive vomiting, diarrhea, or sweating
- · are older than 65 years of age
- are pregnant or think you might be pregnant
- · are breastfeeding

#### INTERACTIONS WITH THIS MEDICATION

As with most medicines, interactions with other drugs are possible. Tell your doctor, nurse, or pharmacist about all the medicines you take, including drugs prescribed by other doctors, vitamins, minerals, natural supplements, or alternative medicines.

IMPORTANT: PLEASE READ

#### Drugs that may interact with Precedex® include:

- anesthestic drugs such as: sevoflurane, isoflurane, propofol, alfentanil, and midazolam
- neuromuscular blockers such as rocuronium, cisatracurium
- · heart medications

#### PROPER USE OF THIS MEDICATION

#### Usual Adult dose:

Dosage will be individualized and titrated to the desired clinical effect. You will be given a loading dose followed by a maintenance dose, specific for your body weight and the procedure you are undergoing. Your doctor will decide what the appropriate dose is for your specific case.

Your doctor and/or nurse will monitor blood pressure, heart rate and oxygen levels, both continuously during the infusion of Precedex<sup>®</sup> and as clinically appropriate after discontinuation.

It is important that following the return of consciousness, you do not attempt to change position or rise from bed without assistance.

### SIDE EFFECTS AND WHAT TO DO ABOUT THEM

You should report symptoms that may occur within 48 hours after you are given Precedex<sup>®</sup> such as: dry mouth, nausea, vomiting, or fever.

#### SERIOUS SIDE EFFECTS, HOW OFTEN THEY HAPPEN AND WHAT TO DO ABOUT THEM

After exposure to Precedex<sup>®</sup>, you should contact your physician or anesthesia professional if you have any of the following reactions:

Symptom / effect

#### Common

Hypotension (low blood pressure): dizziness, fainting, lightheadedness

Hypertension (high blood pressure): headaches, vision disorders, nausea and vomiting

Hyperglycemia (high blood sugar): irregular heartbeats, muscle weakness and generally feeling unwell

Hypokalemia(low potassium blood level): irregular heartbeats, muscle weakness and generally feeling unwell

**Bradycardia**: slow heart beat

Tachycardia: fast heart beat

Hypoxia: blueish colouration to the skin, confusion, fast heartbeat, shortness of breath, sweating Call your doctor immediately or 911.

#### IMPORTANT: PLEASE READ

| Uncommon | |
|---|---|
| Nervousness | Talk with your doctor. |
| Headaches | |
| Agitation | |
| Weakness | |
| Confusion | |
| Excessive sweating | |
| Weight loss | |
| Abdominal pain | |
| Salt cravings | |
| Diarrhea | |
| Constipation | |
| Dizziness/ | |
| Lightheadedness | |
| Anemia: fatigue, loss of | |
| energy, weakness,<br>shortness of breath | |
| | a. !! |
| Respiratory difficulty | Call your doctor immediately or 911. |

This is not a complete list of side effects. For any unexpected effects while taking Precedex<sup>®</sup>, contact your doctor or pharmacist.

#### HOW TO STORE IT

Precedex<sup>®</sup> (100 mcg/mL) is stored between 15 to 30°C.

Precedex<sup>®</sup> (4 mcg/mL) is stored between 15 to 30°C.

Protect from freezing.

#### REPORTING SUSPECTED SIDE EFFECTS

You can report any suspected adverse reactions associated with the use of health products to the Canada Vigilance Program by one of the following 3 ways.

- Report online at <a href="https://www.canada.ca/en/health-canada/services/drugs-health-products/medeffect-canada/adverse-reaction-reporting.html">https://www.canada.ca/en/health-canada/services/drugs-health-products/medeffect-canada/adverse-reaction-reporting.html</a>.
- Call toll-free at 1-866-234-2345
- Complete a Canada Vigilance Reporting Form and:
- Fax toll-free to 1-866-678-6789, or

Mail to: Canada Vigilance Program Health Canada Postal Locator 1908C Ottawa, Ontario K1A 0K9

Postage paid labels, Canada Vigilance Reporting Form and the adverse reaction reporting guidelines are available on the MedEffect<sup>TM</sup> Canada Web site at

https://www.canada.ca/en/health-canada/services/drugs-health products/medeffect-canada/adverse-reaction-reporting.html.

NOTE: Should you require information related to the management of side effects, contact your health professional. The Canada Vigilance Program does not provide medical advice.

#### MORE INFORMATION

This document plus the full product monograph, prepared for health professionals can be found by contacting the sponsor Pfizer Canada Inc. at: 1-800-463-6001.

This leaflet was prepared by: Pfizer Canada Inc. Kirkland, Québec H9J 2M5

Last revised: March 6, 2018